CLINICAL TRIAL: NCT03850483
Title: A PHASE 2B, RANDOMIZED, DOUBLE BLIND, VEHICLE CONTROLLED, PARALLEL-GROUP, DOSE RANGING STUDY TO ASSESS EFFICACY, SAFETY, TOLERABILITY AND PHARMACOKINETICS OF PF-06700841 TOPICAL CREAM APPLIED ONCE OR TWICE DAILY FOR 12 WEEKS IN PARTICIPANTS WITH MILD TO MODERATE CHRONIC PLAQUE PSORIASIS
Brief Title: Dose Ranging Study To Assess Efficacy, Safety and Tolerability Of PF-06700841 Topical Cream In Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7931023; 2018-003051-38 (EudraCT Number)
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Results first posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Psoriasis
Keywords: psoriasis; topical
MeSH Terms: conditions — Psoriasis | interventions — PF-06700841

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Vehicle cream QD (Placebo Comparator): Vehicle cream applied once daily (QD)
  Interventions: Drug: Vehicle (Placebo)
- PF-06700841 0.1% cream QD (Experimental): PF-06700841 0.1% cream applied once daily (QD)
  Interventions: Drug: PF-06700841
- PF-06700841 0.3% cream QD (Experimental): PF-06700841 0.3% cream applied once daily (QD)
  Interventions: Drug: PF-06700841
- PF-06700841 1% cream QD (Experimental): PF-06700841 1% cream applied once daily (QD)
  Interventions: Drug: PF-06700841
- PF-06700841 3% cream QD (Experimental): PF-06700841 3% cream applied once daily (QD)
  Interventions: Drug: PF-06700841
- PF-06700841 0.3% cream BID (Experimental): PF-06700841 0.3% cream applied twice daily (BID)
  Interventions: Drug: PF-06700841
- PF-06700841 1% cream BID (Experimental): PF-06700841 1% cream applied twice daily (BID)
  Interventions: Drug: PF-06700841
- Vehicle cream BID (Placebo Comparator): Vehicle cream applied twice daily (BID)
  Interventions: Drug: Vehicle (Placebo)
- PF-06700841 3% cream BID (Experimental): PF-06700841 3% cream applied twice daily (BID)
  Interventions: Drug: PF-06700841

INTERVENTIONS:
Drug: PF-06700841 — PF-06700841 topical cream
  Arms: PF-06700841 0.1% cream QD; PF-06700841 0.3% cream BID; PF-06700841 0.3% cream QD; PF-06700841 1% cream BID; PF-06700841 1% cream QD; PF-06700841 3% cream BID; PF-06700841 3% cream QD
Drug: Vehicle (Placebo) — Vehicle topical cream
  Arms: Vehicle cream BID; Vehicle cream QD

SUMMARY:
This is a Phase 2b, randomized, double blind, vehicle controlled, parallel group, multicenter study in participants with mild to moderate plaque psoriasis. The duration of study participation will be approximately 22 weeks, including up to a 6 week screening period, 12 week treatment period, and approximately 4 week follow up period. Approximately 280 participants are planned to be randomized into the study.

ELIGIBILITY:
Inclusion Criteria:

* plaque psoriasis for 6 months
* PGA score mild or moderate
* body surface area (BSA) 2-15%

Exclusion Criteria:

* other skin conditions that would interfere with the evaluation of psoriasis
* history of herpes zoster or simplex
* Infected with Mycobacterium tuberculosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (78):
- United States (37):
  - Center for Dermatology and Plastic Surgery/CCT, Scottsdale, Arizona
  - Center for Dermatology and Plastic Surgery, Scottsdale, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - California Skin Institute, Anaheim, California
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - First OC Dermatology, Fountain Valley, California
  - Clinical Science Institute, Santa Monica, California
  - New England Research Associates, LLC, Bridgeport, Connecticut
  - Dermatology Physicians of Connecticut, Shelton, Connecticut
  - Olympian Clinical Research, Clearwater, Florida
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Renstar Medical Research, Ocala, Florida
  - MidState Skin Institute, Ocala, Florida
  - Park Avenue Dermatology, PA, Orange Park, Florida
  - Center for Clinical Studies, Tampa, Florida
  - Dundee Dermatology, West Dundee, Illinois
  - Ds Research, Clarksville, Indiana
  - DS Research, Louisville, Kentucky
  - Meridian Clinical Research, LLC, Baton Rouge, Louisiana
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Hassman Research Institute, Berlin, New Jersey
  - Psoriasis Treatment Center of Central New Jersey, East Windsor, New Jersey
  - Bayside Dermatology Center, Bayside, New York
  - Dermatology Consulting Services, PLLC, High Point, North Carolina
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Vital Prospects Clinical Research Institute, PC, Tulsa, Oklahoma
  - Health Concepts, Rapid City, South Dakota
  - Rivergate Dermatology Clinical Research, Goodlettsville, Tennessee
  - Austin Institute for Clinical Research, Inc., Austin, Texas
  - studies in Dermatology, LLC, Cypress, Texas
  - Center for Clinical Studies, LTD. LLP, Houston, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Center for Clinical Studies, Webster, Texas
  - Summit Clinical Research, LLC, Franklin, Virginia
  - Virginia Dermatology and Skin Cancer Center, Norfolk, Virginia
- Australia (4):
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Emeritus Research, Camberwell, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - Cabrini Hospital, Malvern, Victoria
- Bulgaria (4):
  - Center for Skin and Venereal Diseases EOOD - Sofia, Sofia
  - DCC Alexandrovska, Sofia
  - Diagnostic Consultative Center - Fokus-5 - Medical Establishment for Outpatient Care OOD, Sofia
  - Dermatological Clinic Sofia, Sofia
- Canada (4):
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - SKiN Health, Cobourg, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
- Gentofte Hospital, Hellerup, Denmark
- Germany (10):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Emovis GmbH, Berlin
  - Rothhaar Studien GmbH, Berlin
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Klinikum Bielefeld gem.GmbH, Bielefeld
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - MENSINGDERMA research GmbH, Hamburg
  - MVZ Alstermed GmbH, Hamburg
  - Dermatologische Gemeinschaftspraxis, Mahlow
  - Klinische Forschung Schwerin GmbH, Schwerin
- Hungary (4):
  - Semmelweis Egyetem Altalanos Orvostudomanyi Kar, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bacs-Kiskun Megyei Korhaz Szegedi Tudomanyegyetem Altalanos Orvostudomanyi Kar Oktato Korhaza, Kecskemét
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Japan (6):
  - Kitago Dermatology Clinic, Sapporo, Hokkaido
  - Nakatsuhifuka Clinic, Kita-ku, Osaka-shi, Osaka
  - Parkside Hiroo Ladies Clinic, Minato-ku, Tokyo
  - Tanpopo Skin Clinic, Ōta-ku, Tokyo
  - Samoncho Dermatological Clinic, Shinjuku-ku, Tokyo
  - Medical Corporation Jitai-kai Tachikawa Dermatology Clinic, Tachikawa, Tokyo
- Latvia (4):
  - Riga 1st Hospital, Riga
  - Aesthetic dermatology clinic of Prof. J. Kisis, Riga
  - Health and Aesthetics Ltd, Riga
  - Outpatient Clinic of Ventspils, Ventspils
- Poland (4):
  - Zdrowie Osteo-Medic s.c. LiA Racewicz, AiJ Supronik, Bialystok
  - Nasz Lekarz Przychodnie Medyczne, Torun
  - MTZ Clinical Research Sp. z o.o, Warsaw
  - WroMedica I. Bielicka, A. Strzalkowska s.c., Wroclaw

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Background] Forman SB, Pariser DM, Poulin Y, Vincent MS, Gilbert SA, Kieras EM, Qiu R, Yu D, Papacharalambous J, Tehlirian C, Peeva E. TYK2/JAK1 Inhibitor PF-06700841 in Patients with Plaque Psoriasis: Phase IIa, Randomized, Double-Blind, Placebo-Controlled Trial. J Invest Dermatol. 2020 Dec;140(12):2359-2370.e5. doi: 10.1016/j.jid.2020.03.962. Epub 2020 Apr 18. PMID 32311398
- [Derived] Draelos ZD, Bushmakin AG, Ghosh P, Xenakis J, Cappelleri JC. Validation of the Peak Pruritus-Numerical Rating Scale in patients with chronic plaque psoriasis: results from a phase 2 study. Int J Dermatol. 2024 Dec;63(12):e375-e382. doi: 10.1111/ijd.17428. Epub 2024 Aug 19. PMID 39160651
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7931023

RESULTS

PARTICIPANT FLOW:
Groups:
- Stage 1: Vehicle Once Daily (QD): During stage 1 of the study participants topically applied vehicle cream on psoriatic areas QD for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- Stage 1: PF-06700841 0.1% QD: During stage 1 of the study participants topically applied PF-06700841 0.1 percent (%) cream on psoriatic areas QD for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- Stage 1: PF-06700841 0.3% QD: During stage 1 of the study participants topically applied PF-06700841 0.3% cream on psoriatic areas QD for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- Stage 1: PF-06700841 1.0% QD: During stage 1 of the study participants topically applied PF-06700841 1.0% cream on psoriatic areas QD for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- Stage 1: PF-06700841 3.0% QD: During stage 1 of the study participants topically applied PF-06700841 3.0% cream on psoriatic areas QD for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- Stage 1: Vehicle Twice Daily (BID): During stage 1 of the study participants topically applied vehicle cream on psoriatic areas BID for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- Stage 1: PF-06700841 0.3% BID: During stage 1 of the study participants topically applied PF-06700841 0.3% cream on psoriatic areas BID for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- Stage 1: PF-06700841 1.0% BID: During stage 1 of the study participants topically applied PF-06700841 1.0% cream on psoriatic areas BID for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- Stage 2: Vehicle BID: During stage 2 of the study participants topically applied vehicle cream on psoriatic areas BID for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- Stage 2: PF-06700841 3.0% BID: During stage 2 of the study participants topically applied PF-06700841 3.0% cream on psoriatic areas BID for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
Period: Treatment for Stage 1
Arm/Group | Stage 1: Vehicle Once Daily (QD) | Stage 1: PF-06700841 0.1% QD | Stage 1: PF-06700841 0.3% QD | Stage 1: PF-06700841 1.0% QD | Stage 1: PF-06700841 3.0% QD | Stage 1: Vehicle Twice Daily (BID) | Stage 1: PF-06700841 0.3% BID | Stage 1: PF-06700841 1.0% BID | Stage 2: Vehicle BID | Stage 2: PF-06700841 3.0% BID
Started | 37 | 37 | 37 | 36 | 37 | 38 | 36 | 36 | 0 | 0
Treated | 37 | 37 | 37 | 36 | 37 | 37 | 36 | 36 | 0 | 0
Completed | 29 | 29 | 26 | 30 | 28 | 27 | 25 | 30 | 0 | 0
Not Completed | 8 | 8 | 11 | 6 | 9 | 11 | 11 | 6 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 3 | 0 | 2 | 0 | 2 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 2 | 2 | 2 | 1 | 2 | 3 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Non-Compliance With Study Drug | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — No Longer Met Eligibility Criteria | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 2 | 3 | 2 | 4 | 3 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Refused Further Treatment | 1 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Randomized but not Treated | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Follow-up for Stage 1
Arm/Group | Stage 1: Vehicle Once Daily (QD) | Stage 1: PF-06700841 0.1% QD | Stage 1: PF-06700841 0.3% QD | Stage 1: PF-06700841 1.0% QD | Stage 1: PF-06700841 3.0% QD | Stage 1: Vehicle Twice Daily (BID) | Stage 1: PF-06700841 0.3% BID | Stage 1: PF-06700841 1.0% BID | Stage 2: Vehicle BID | Stage 2: PF-06700841 3.0% BID
Started | 37 | 37 | 37 | 36 | 37 | 37 | 36 | 36 | 0 | 0
Completed | 37 | 34 | 35 | 34 | 34 | 33 | 34 | 33 | 0 | 0
Not Completed | 0 | 3 | 2 | 2 | 3 | 4 | 2 | 3 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Refused Further Study Procedures | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 2 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Period: Treatment for Stage 2
Arm/Group | Stage 1: Vehicle Once Daily (QD) | Stage 1: PF-06700841 0.1% QD | Stage 1: PF-06700841 0.3% QD | Stage 1: PF-06700841 1.0% QD | Stage 1: PF-06700841 3.0% QD | Stage 1: Vehicle Twice Daily (BID) | Stage 1: PF-06700841 0.3% BID | Stage 1: PF-06700841 1.0% BID | Stage 2: Vehicle BID | Stage 2: PF-06700841 3.0% BID
Started | 0 (Stage 1 enrolment was different from Stage 2.) | 0 (Stage 1 enrolment was different from Stage 2.) | 0 (Stage 1 enrolment was different from Stage 2.) | 0 (Stage 1 enrolment was different from Stage 2.) | 0 (Stage 1 enrolment was different from Stage 2.) | 0 (Stage 1 enrolment was different from Stage 2.) | 0 (Stage 1 enrolment was different from Stage 2.) | 0 (Stage 1 enrolment was different from Stage 2.) | 12 (Stage 1 enrolment was different from Stage 2.) | 38 (Stage 1 enrolment was different from Stage 2.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 27
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 5
Not completed — No Longer Meets Eligibility Criteria | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Refused Further Treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Follow-up For Stage 2
Arm/Group | Stage 1: Vehicle Once Daily (QD) | Stage 1: PF-06700841 0.1% QD | Stage 1: PF-06700841 0.3% QD | Stage 1: PF-06700841 1.0% QD | Stage 1: PF-06700841 3.0% QD | Stage 1: Vehicle Twice Daily (BID) | Stage 1: PF-06700841 0.3% BID | Stage 1: PF-06700841 1.0% BID | Stage 2: Vehicle BID | Stage 2: PF-06700841 3.0% BID
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 38
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 36
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis population included participants who were randomly assigned to PF-06700841 and applied at least 1 dose of PF-06700841.
Groups:
- Vehicle Once Daily (QD): During stage 1 of the study participants topically applied vehicle cream on psoriatic areas QD for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- PF-06700841 0.1% QD: During stage 1 of the study participants topically applied PF-06700841 0.1% cream on psoriatic areas QD for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- PF-06700841 0.3% QD: During stage 1 of the study participants topically applied PF-06700841 0.3% cream on psoriatic areas QD for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- PF-06700841 1.0% QD: During stage 1 of the study participants topically applied PF-06700841 1.0% cream on psoriatic areas QD for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- PF-06700841 3.0% QD: During stage 1 of the study participants topically applied PF-06700841 3.0% cream on psoriatic areas QD for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- Pooled Vehicle BID: During stage 1 and 2 of the study participants topically applied vehicle cream on psoriatic areas BID for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- PF-06700841 0.3% BID: During stage 1 of the study participants topically applied PF-06700841 0.3% cream on psoriatic areas BID for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- PF-06700841 1.0% BID: During stage 1 of the study participants topically applied PF-06700841 1.0% cream on psoriatic areas BID for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- PF-06700841 3.0% BID: During stage 2 of the study participants topically applied PF-06700841 3.0% cream on psoriatic areas BID for a maximum of 12 weeks. Participants were followed up for 4 weeks after last dose.
- Total: Total of all reporting groups
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID | Total
Number analyzed (Participants) | 37 | 37 | 37 | 36 | 37 | 49 | 36 | 36 | 38 | 343
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.6 (15.83) | 51.8 (12.49) | 51.4 (12.26) | 49.4 (15.30) | 48.4 (12.37) | 50.9 (12.85) | 48.2 (13.58) | 50.9 (16.45) | 48.9 (12.93) | 49.9 (13.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 7 | 6 | 13 | 18 | 11 | 11 | 14 | 102
  Male | 25 | 27 | 30 | 30 | 24 | 31 | 25 | 25 | 24 | 241
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 4 | 1 | 2 | 8 | 3 | 3 | 7 | 35
  Not Hispanic or Latino | 32 | 35 | 33 | 35 | 35 | 39 | 33 | 33 | 31 | 306
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Asian | 6 | 4 | 6 | 6 | 4 | 3 | 6 | 3 | 2 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 2 | 7
  White | 30 | 33 | 28 | 30 | 32 | 45 | 30 | 31 | 34 | 293
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Week 12
Description: The Psoriasis Area and Severity Index (PASI) score (0-72, with higher score representing greater severity) is a measurement of the severity and extent of psoriasis. The four regions of the body parts are head (10%), arms (20%), trunk (30%) and legs (40%). In each region, the area is expressed as a score of 0 (nothing), 1 (1-9%), 2 (10-29%), 3 (30-49%), 4 (50-69%), 5 (70-89%) or 6 (90-100%). Within each area, the degree of severity for erythema, induration and scaling are estimated between 0 and 4, with 4 being the highest severity. The final score combines disease severity and effected body surface area (BSA) from for four regions using the formula PASI =0.1Ah(Eh + Ih + Sh) + 0.2Au(Eu + Iu + Su) + 0.3At(Et + It + St) + 0.4Al(El + Il + Sl) where A = Area Score; E = erythema; I =induration; S = scaling; h = head; u = upper limbs; t = trunk; l = lower limbs.
Time Frame: Baseline, Week 12
Population: Efficacy analysis set (EAS) included all randomized participants who receive at least 1 dose of investigational product (PF-06700841 or placebo) and Week 12 visits were not missing due to COVID-19 pandemic.
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 36 | 37 | 37 | 36 | 37 | 49 | 36 | 35 | 38
Unit on a scale | -1.6 (0.46) | -2.2 (0.46) | -1.4 (0.46) | -2.2 (0.46) | -2.4 (0.45) | -2.2 (0.42) | -2.5 (0.53) | -3.0 (0.51) | -2.8 (0.48)
Statistical Analysis 1: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Test type: Superiority; p = 0.1641, ANCOVA — Multiplicity adjustment comparing 6 different treatment arms was performed only for the primary endpoint using Hochberg step-up procedure to maintain overall familywise error rate at 5% level; Least square (LS) mean difference = -0.6, 90% CI 2-sided [-1.71 to 0.43], Standard Error of Mean 0.65
Statistical Analysis 2: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Test type: Superiority; p = 0.6100, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 0.2, 90% CI 2-sided [-0.89 to 1.26], Standard Error of Mean 0.65
Statistical Analysis 3: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Test type: Superiority; p = 0.1686, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -0.6, 90% CI 2-sided [-1.70 to 0.45], Standard Error of Mean 0.65
Statistical Analysis 4: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Test type: Superiority; p = 0.1051, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -0.8, 90% CI 2-sided [-1.87 to 0.25], Standard Error of Mean 0.64
Statistical Analysis 5: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Test type: Superiority; p = 0.3583, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -0.2, 90% CI 2-sided [-1.37 to 0.88], Standard Error of Mean 0.68
Statistical Analysis 6: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Test type: Superiority; p = 0.1131, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -0.8, 90% CI 2-sided [-1.88 to 0.29], Standard Error of Mean 0.66
Statistical Analysis 7: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Test type: Superiority; p = 0.1812, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -0.6, 90% CI 2-sided [-1.64 to 0.47], Standard Error of Mean 0.64

2. Secondary Outcome: Percentage of Participants With Physician Global Assessment (PGA) Score Clear (0) or Almost Clear (1) and Greater Than or Equal to (>=) 2 Points Improvement From Baseline at Week 12
Description: PGA of psoriasis was scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling were scored separately over the whole body according to a 5-point severity scale (0 [no symptom] to 4 [severe symptom]). The total score was calculated as average of the 3 severity scores and rounded to the nearest whole number score to determine the PGA score and category. Scale for PGA: 0= clear, 1= almost clear, 2= mild, 3= moderate and 4= severe. Higher scores indicate more severity.
Time Frame: Baseline, Week 12
Population: EAS included all randomized participants who receive at least 1 dose of investigational product (PF-06700841 or placebo) and Week 12 visits were not missing due to COVID-19 pandemic. Here, 'overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 29 | 29 | 26 | 29 | 28 | 34 | 24 | 29 | 28
Percentage of participants | 6.9 [1.8 to 20.0] | 10.3 [3.9 to 22.9] | 15.4 [6.9 to 29.9] | 10.3 [3.9 to 22.9] | 21.4 [9.8 to 36.6] | 14.7 [7.3 to 26.9] | 20.8 [10.5 to 37.0] | 27.6 [14.5 to 42.5] | 17.9 [8.9 to 33.3]
Statistical Analysis 1: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Test type: Superiority; p = 0.3747, Chan and Zhang method; Risk Difference (RD) = 3.4, 90% CI 2-sided [-10.6 to 17.9]
Statistical Analysis 2: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Test type: Superiority; p = 0.2430, Chan and Zhang method; Risk Difference (RD) = 8.5, 90% CI 2-sided [-6.6 to 25.9]
Statistical Analysis 3: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Test type: Superiority; p = 0.3747, Chan and Zhang method; Risk Difference (RD) = 3.4, 90% CI 2-sided [-10.6 to 17.9]
Statistical Analysis 4: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Test type: Superiority; p = 0.0665, Chan and Zhang method; Risk Difference (RD) = 14.5, 0.0665% CI 2-sided [-1.3 to 31.5]
Statistical Analysis 5: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Test type: Superiority; p = 0.3423, Chan and Zhang method; Risk Difference (RD) = 6.1, 90% CI 2-sided [-12.1 to 25.5]
Statistical Analysis 6: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Test type: Superiority; p = 0.1271, Chan and Zhang method; Risk Difference (RD) = 12.9, 90% CI 2-sided [-4.7 to 30.9]
Statistical Analysis 7: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Test type: Superiority; p = 0.4010, Chan and Zhang method; Risk Difference (RD) = 3.2, 90% CI 2-sided [-13.2 to 21.1]

3. Secondary Outcome: Percentage of Participants With 75% Reduction From Baseline in PASI at Week 1, 2, 4, 6, 8, 10, 12, 14, and 16
Description: The PASI score (0-72, with higher score representing greater severity) is a measurement of the severity and extent of psoriasis. The four regions of the body parts are head (10%), arms (20%), trunk (30%) and legs (40%). In each region, the area is expressed as a score of 0 (nothing), 1 (1-9%), 2 (10-29%), 3 (30-49%), 4 (50-69%), 5 (70-89%) or 6 (90-100%). Within each area, the degree of severity for erythema, induration and scaling are estimated between 0 and 4, with 4 being the highest severity. The final score combines disease severity and effected BSA from for four regions using the formula PASI =0.1Ah(Eh + Ih + Sh) + 0.2Au(Eu + Iu + Su) + 0.3At(Et + It + St) + 0.4Al(El + Il + Sl) where A = Area Score; E = erythema; I =induration; S = scaling; h = head; u = upper limbs; t = trunk; l = lower limbs.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10, 12, 14, and 16
Population: EAS included all randomized participants who receive at least 1 dose of investigational product (PF-06700841 or placebo) and Week 12 visits were not missing due to COVID-19 pandemic. Here, 'overall number of participants analyzed' signifies number of participants evaluable for this outcome measure and 'number analyzed' signifies number of participants evaluable at specified time points.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 32 | 36 | 34 | 35 | 35 | 45 | 35 | 34 | 37
Percentage of participants
  Week 1: number analyzed (Participants) | 32 | 33 | 34 | 35 | 35 | 45 | 32 | 34 | 37
  Week 1 | 3.1 [0.3 to 13.1] | 3.0 [0.3 to 12.7] | 0 [0.0 to 8.0] | 0 [0.0 to 7.7] | 0 [0.0 to 7.7] | 0 [0.0 to 6.0] | 0 [0.0 to 8.5] | 2.9 [0.3 to 12.3] | 2.7 [0.3 to 11.2]
  Week 2: number analyzed (Participants) | 32 | 36 | 31 | 35 | 35 | 45 | 35 | 32 | 35
  Week 2 | 3.1 [0.3 to 13.1] | 0 [0.0 to 7.5] | 0 [0.0 to 8.8] | 2.9 [0.3 to 11.9] | 0 [0.0 to 7.7] | 2.2 [0.2 to 9.2] | 0 [0.0 to 7.7] | 6.3 [1.7 to 18.0] | 5.7 [1.5 to 16.4]
  week 4: number analyzed (Participants) | 32 | 32 | 28 | 34 | 34 | 45 | 30 | 33 | 33
  week 4 | 3.1 [0.3 to 13.1] | 0 [0.0 to 8.5] | 3.6 [0.4 to 15.1] | 0 [0.0 to 8.0] | 0 [0.0 to 8.0] | 8.9 [3.9 to 18.0] | 6.7 [1.8 to 19.3] | 3.0 [0.3 to 12.7] | 12.1 [5.4 to 25.1]
  Week 6: number analyzed (Participants) | 31 | 31 | 27 | 31 | 29 | 36 | 28 | 28 | 29
  Week 6 | 3.2 [0.3 to 13.5] | 0 [0.0 to 8.8] | 7.4 [2.0 to 20.4] | 6.5 [1.7 to 18.7] | 10.3 [3.9 to 22.9] | 13.9 [6.9 to 25.4] | 10.7 [4.0 to 23.8] | 10.7 [4.0 to 23.8] | 10.3 [3.9 to 22.9]
  Week 8: number analyzed (Participants) | 30 | 30 | 27 | 31 | 28 | 36 | 25 | 29 | 28
  Week 8 | 6.7 [1.8 to 19.3] | 6.7 [1.8 to 19.3] | 7.4 [2.0 to 20.4] | 6.5 [1.7 to 18.7] | 14.3 [6.4 to 28.4] | 13.9 [6.9 to 25.4] | 16.0 [7.2 to 30.7] | 13.8 [6.2 to 27.9] | 14.3 [6.4 to 28.4]
  Week 10: number analyzed (Participants) | 29 | 30 | 25 | 29 | 28 | 33 | 24 | 28 | 26
  Week 10 | 10.3 [3.9 to 22.9] | 3.3 [0.4 to 14.0] | 8.0 [2.1 to 21.4] | 17.2 [8.6 to 32.0] | 14.3 [6.4 to 28.4] | 18.2 [8.2 to 31.3] | 20.8 [10.5 to 37.0] | 10.7 [4.0 to 23.8] | 15.4 [6.9 to 29.9]
  Week 12: number analyzed (Participants) | 29 | 29 | 26 | 29 | 28 | 34 | 24 | 29 | 28
  Week 12 | 10.3 [3.9 to 22.9] | 10.3 [3.9 to 22.9] | 7.7 [2.1 to 20.9] | 20.7 [9.4 to 35.2] | 17.9 [8.9 to 33.3] | 20.6 [11.3 to 34.9] | 12.5 [4.7 to 28.2] | 24.1 [13.4 to 38.5] | 17.9 [8.9 to 33.3]
  Week 14: number analyzed (Participants) | 29 | 26 | 23 | 28 | 28 | 29 | 23 | 25 | 27
  Week 14 | 3.4 [0.4 to 14.5] | 7.7 [2.1 to 20.9] | 8.7 [2.3 to 22.8] | 21.4 [9.8 to 36.6] | 14.3 [6.4 to 28.4] | 10.3 [3.9 to 22.9] | 13.0 [4.9 to 29.6] | 20.0 [10.1 to 36.2] | 14.8 [6.6 to 29.1]
  Week 16: number analyzed (Participants) | 29 | 27 | 23 | 28 | 26 | 31 | 23 | 24 | 26
  Week 16 | 3.4 [0.4 to 14.5] | 11.1 [4.2 to 24.8] | 17.4 [7.8 to 33.5] | 25.0 [13.9 to 40.0] | 15.4 [6.9 to 29.9] | 16.1 [8.1 to 29.7] | 13.0 [4.9 to 29.6] | 12.5 [4.7 to 28.2] | 15.4 [6.9 to 29.9]
Statistical Analysis 1: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 1; Test type: Superiority; p = 0.4225, Chan and Zhang method; Risk Difference (RD) = -0.1, 90% CI 2-sided [-11.2 to 10.4]
Statistical Analysis 2: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 1; Test type: Superiority; p = 0.7483, Chan and Zhang method; Risk Difference (RD) = -3.1, 90% CI 2-sided [-14.0 to 5.0]
Statistical Analysis 3: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 1; Test type: Superiority; p = 0.7539, Chan and Zhang method; Risk Difference (RD) = -3.1, 90% CI 2-sided [-14.0 to 4.8]
Statistical Analysis 4: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 1; Test type: Superiority; p = 0.7539, Chan and Zhang method; Risk Difference (RD) = -3.1, 90% CI 2-sided [-14.0 to 4.8]
Statistical Analysis 5: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 1; Test type: Superiority; p = 0.5000, Chan and Zhang method; Risk Difference (RD) = 0.0, 90% CI 2-sided [-6.4 to 8.9]
Statistical Analysis 6: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 1; Test type: Superiority; p = 0.2125, Chan and Zhang method; Risk Difference (RD) = 2.9, 90% CI 2-sided [-3.4 to 13.2]
Statistical Analysis 7: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 1; Test type: Superiority; p = 0.2267, Chan and Zhang method; Risk Difference (RD) = 2.7, 90% CI 2-sided [-3.5 to 12.2]
Statistical Analysis 8: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 2; Test type: Superiority; p = 0.7592, Chan and Zhang method; Risk Difference (RD) = -3.1, 90% CI 2-sided [-14.0 to 4.6]
Statistical Analysis 9: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 2; Test type: Superiority; p = 0.7299, Chan and Zhang method; Risk Difference (RD) = -3.1, 90% CI 2-sided [-14.0 to 5.5]
Statistical Analysis 10: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 2; Test type: Superiority; p = 0.4463, Chan and Zhang method; Risk Difference (RD) = -0.3, 90% CI 2-sided [-11.3 to 9.4]
Statistical Analysis 11: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 2; Test type: Superiority; p = 0.7539, Chan and Zhang method; Risk Difference (RD) = -3.1, 90% CI 2-sided [-14.0 to 4.8]
Statistical Analysis 12: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 2; Test type: Superiority; p = 0.7009, Chan and Zhang method; Risk Difference (RD) = -2.2, 90% CI 2-sided [-10.1 to 5.9]
Statistical Analysis 13: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 2; Test type: Superiority; p = 0.2507, Chan and Zhang method; Risk Difference (RD) = 4.0, 90% CI 2-sided [-4.5 to 15.6]
Statistical Analysis 14: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 2; Test type: Superiority; p = 0.2993, Chan and Zhang method; Risk Difference (RD) = 3.5, 90% CI 2-sided [-4.8 to 14.3]
Statistical Analysis 15: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 4; Test type: Superiority; p = 0.7363, Chan and Zhang method; Risk Difference (RD) = -3.1, 90% CI 2-sided [-14.0 to 5.5]
Statistical Analysis 16: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 4; Test type: Superiority; p = 0.5369, Chan and Zhang method; Risk Difference (RD) = 0.4, 90% CI 2-sided [-10.5 to 12.3]
Statistical Analysis 17: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 4; Test type: Superiority; p = 0.7483, Chan and Zhang method; Risk Difference (RD) = -3.1, 90% CI 2-sided [-14.0 to 5.0]
Statistical Analysis 18: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 4; Test type: Superiority; p = 0.7483, Chan and Zhang method; Risk Difference (RD) = -3.1, 90% CI 2-sided [-14.0 to 5.0]
Statistical Analysis 19: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 4; Test type: Superiority; p = 0.5990, Chan and Zhang method; Risk Difference (RD) = -2.2, 90% CI 2-sided [-13.7 to 11.6]
Statistical Analysis 20: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 4; Test type: Superiority; p = 0.7926, Chan and Zhang method; Risk Difference (RD) = -5.9, 90% CI 2-sided [-16.4 to 4.9]
Statistical Analysis 21: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 4; Test type: Superiority; p = 0.3402, Chan and Zhang method; Risk Difference (RD) = 3.2, 90% CI 2-sided [-9.0 to 17.6]
Statistical Analysis 22: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 6; Test type: Superiority; p = 0.7364, Chan and Zhang method; Risk Difference (RD) = -3.2, 90% CI 2-sided [-14.4 to 5.7]
Statistical Analysis 23: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 6; Test type: Superiority; p = 0.3009, Chan and Zhang method; Risk Difference (RD) = 4.2, 90% CI 2-sided [-7.4 to 17.7]
Statistical Analysis 24: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 6; Test type: Superiority; p = 0.3400, Chan and Zhang method; Risk Difference (RD) = 3.2, 90% CI 2-sided [-8.1 to 15.9]
Statistical Analysis 25: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 6; Test type: Superiority; p = 0.1631, Chan and Zhang method; Risk Difference (RD) = 7.1, 90% CI 2-sided [-4.8 to 21.1]
Statistical Analysis 26: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 6; Test type: Superiority; p = 0.6214, Chan and Zhang method; Risk Difference (RD) = -3.2, 90% CI 2-sided [-17.8 to 13.0]
Statistical Analysis 27: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 6; Test type: Superiority; p = 0.6214, Chan and Zhang method; Risk Difference (RD) = -3.2, 90% CI 2-sided [-17.8 to 13.0]
Statistical Analysis 28: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 6; Test type: Superiority; p = 0.6413, Chan and Zhang method; Risk Difference (RD) = -3.5, 90% CI 2-sided [-17.9 to 11.7]
Statistical Analysis 29: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 8; Test type: Superiority; p = 0.5000, Chan and Zhang method; Risk Difference (RD) = 0.0, 90% CI 2-sided [-13.1 to 13.1]
Statistical Analysis 30: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 8; Test type: Superiority; p = 0.5134, Chan and Zhang method; Risk Difference (RD) = 0.7, 90% CI 2-sided [-12.6 to 15.2]
Statistical Analysis 31: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 8; Test type: Superiority; p = 0.4468, Chan and Zhang method; Risk Difference (RD) = -0.2, 90% CI 2-sided [-13.4 to 12.5]
Statistical Analysis 32: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 8; Test type: Superiority; p = 0.2778, Chan and Zhang method; Risk Difference (RD) = 7.6, 90% CI 2-sided [-6.8 to 23.9]
Statistical Analysis 33: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 8; Test type: Superiority; p = 0.4571, Chan and Zhang method; Risk Difference (RD) = 2.1, 90% CI 2-sided [-14.5 to 21.0]
Statistical Analysis 34: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 8; Test type: Superiority; p = 0.4741, Chan and Zhang method; Risk Difference (RD) = -0.1, 90% CI 2-sided [-15.3 to 16.7]
Statistical Analysis 35: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 8; Test type: Superiority; p = 0.5153, Chan and Zhang method; Risk Difference (RD) = 0.4, 90% CI 2-sided [-14.8 to 16.7]
Statistical Analysis 36: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 10; Test type: Superiority; p = 0.8287, Chan and Zhang method; Risk Difference (RD) = -7.0, 90% CI 2-sided [-21.1 to 5.3]
Statistical Analysis 37: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 10; Test type: Superiority; p = 0.5675, Chan and Zhang method; Risk Difference (RD) = -2.3, 90% CI 2-sided [-17.8 to 14.2]
Statistical Analysis 38: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 10; Test type: Superiority; p = 0.2648, Chan and Zhang method; Risk Difference (RD) = 6.9, 90% CI 2-sided [-9.8 to 23.2]
Statistical Analysis 39: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 10; Test type: Superiority; p = 0.3792, Chan and Zhang method; Risk Difference (RD) = 3.9, 90% CI 2-sided [-11.8 to 20.8]
Statistical Analysis 40: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 10; Test type: Superiority; p = 0.4438, Chan and Zhang method; Risk Difference (RD) = 2.7, 90% CI 2-sided [-16.3 to 23.1]
Statistical Analysis 41: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 10; Test type: Superiority; p = 0.7014, Chan and Zhang method; Risk Difference (RD) = -7.5, 90% CI 2-sided [-23.3 to 9.4]
Statistical Analysis 42: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 10; Test type: Superiority; p = 0.5841, Chan and Zhang method; Risk Difference (RD) = -2.8, 90% CI 2-sided [-19.7 to 15.0]
Statistical Analysis 43: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 12; Test type: Superiority; p = 0.5000, Chan and Zhang method; Risk Difference (RD) = 0.0, 90% CI 2-sided [-15.3 to 15.3]
Statistical Analysis 44: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 12; Test type: Superiority; p = 0.5834, Chan and Zhang method; Risk Difference (RD) = -2.7, 90% CI 2-sided [-17.5 to 12.3]
Statistical Analysis 45: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 12; Test type: Superiority; p = 0.1534, Chan and Zhang method; Risk Difference (RD) = 10.3, 90% CI 2-sided [-6.4 to 27.2]
Statistical Analysis 46: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 12; Test type: Superiority; p = 0.2720, Chan and Zhang method; Risk Difference (RD) = 7.5, 90% CI 2-sided [-8.8 to 24.9]
Statistical Analysis 47: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 12; Test type: Superiority; p = 0.6815, Chan and Zhang method; Risk Difference (RD) = -8.1, 90% CI 2-sided [-25.1 to 10.4]
Statistical Analysis 48: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 12; Test type: Superiority; p = 0.3900, Chan and Zhang method; Risk Difference (RD) = 3.5, 90% CI 2-sided [-14.4 to 22.0]
Statistical Analysis 49: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 12; Test type: Superiority; p = 0.5865, Chan and Zhang method; Risk Difference (RD) = -2.7, 90% CI 2-sided [-20.0 to 15.9]
Statistical Analysis 50: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 14; Test type: Superiority; p = 0.3087, Chan and Zhang method; Risk Difference (RD) = 4.2, 90% CI 2-sided [-8.2 to 18.9]
Statistical Analysis 51: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 14; Test type: Superiority; p = 0.3137, Chan and Zhang method; Risk Difference (RD) = 5.2, 90% CI 2-sided [-8.2 to 20.9]
Statistical Analysis 52: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 14; Test type: Superiority; p = 0.0245, Chan and Zhang method; Risk Difference (RD) = 18.0, 90% CI 2-sided [2.7 to 34.8]
Statistical Analysis 53: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 14; Test type: Superiority; p = 0.1119, Chan and Zhang method; Risk Difference (RD) = 10.8, 90% CI 2-sided [-3.0 to 26.0]
Statistical Analysis 54: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 14; Test type: Superiority; p = 0.4140, Chan and Zhang method; Risk Difference (RD) = 2.7, 90% CI 2-sided [-13.2 to 20.4]
Statistical Analysis 55: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 14; Test type: Superiority; p = 0.2356, Chan and Zhang method; Risk Difference (RD) = 9.7, 90% CI 2-sided [-7.2 to 28.5]
Statistical Analysis 56: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 14; Test type: Superiority; p = 0.3638, Chan and Zhang method; Risk Difference (RD) = 4.5, 90% CI 2-sided [-11.5 to 21.5]
Statistical Analysis 57: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 16; Test type: Superiority; p = 0.1613, Chan and Zhang method; Risk Difference (RD) = 7.7, 90% CI 2-sided [-5.2 to 22.9]
Statistical Analysis 58: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 16; Test type: Superiority; p = 0.0557, Chan and Zhang method; Risk Difference (RD) = 13.9, 90% CI 2-sided [-0.5 to 31.4]
Statistical Analysis 59: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 16; Test type: Superiority; p = 0.0114, Chan and Zhang method; Risk Difference (RD) = 21.6, 90% CI 2-sided [5.6 to 38.3]
Statistical Analysis 60: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 16; Test type: Superiority; p = 0.0753, Chan and Zhang method; Risk Difference (RD) = 11.9, 90% CI 2-sided [-1.8 to 28.1]
Statistical Analysis 61: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 16; Test type: Superiority; p = 0.5635, Chan and Zhang method; Risk Difference (RD) = -3.1, 90% CI 2-sided [-20.1 to 15.2]
Statistical Analysis 62: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 16; Test type: Superiority; p = 0.6201, Chan and Zhang method; Risk Difference (RD) = -3.6, 90% CI 2-sided [-20.3 to 14.5]
Statistical Analysis 63: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 16; Test type: Superiority; p = 0.4792, Chan and Zhang method; Risk Difference (RD) = -0.7, 90% CI 2-sided [-17.6 to 17.0]

4. Secondary Outcome: Change From Baseline in PASI Scores at Week 1, 2, 4, 6, 8, 10 and 12
Description: as for outcome 3
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 32 | 36 | 34 | 35 | 35 | 45 | 35 | 34 | 37
Unit on a scale
  Change at Week 1: number analyzed (Participants) | 32 | 33 | 34 | 35 | 35 | 45 | 32 | 34 | 37
  Change at Week 1 | -0.9 (0.22) | -0.7 (0.22) | -0.6 (0.22) | -0.9 (0.22) | -0.8 (0.22) | -0.5 (0.19) | -0.7 (0.23) | -0.7 (0.22) | -0.8 (0.22)
  Change at Week 2: number analyzed (Participants) | 32 | 36 | 31 | 35 | 35 | 45 | 35 | 32 | 35
  Change at Week 2 | -1.4 (0.26) | -0.7 (0.26) | -0.9 (0.27) | -1.4 (0.26) | -1.3 (0.26) | -0.8 (0.25) | -1.4 (0.29) | -1.6 (0.29) | -1.7 (0.29)
  Change at Week 4: number analyzed (Participants) | 32 | 32 | 28 | 34 | 34 | 45 | 30 | 33 | 33
  Change at Week 4 | -1.4 (0.31) | -1.2 (0.31) | -1.2 (0.33) | -1.4 (0.31) | -1.6 (0.31) | -1.0 (0.35) | -2.3 (0.42) | -1.7 (0.41) | -2.2 (0.41)
  Change at Week 6: number analyzed (Participants) | 31 | 31 | 27 | 31 | 29 | 36 | 28 | 28 | 29
  Change at Week 6 | -1.5 (0.35) | -1.4 (0.35) | -1.2 (0.37) | -1.6 (0.35) | -2.4 (0.36) | -1.2 (0.37) | -2.5 (0.45) | -2.1 (0.44) | -2.1 (0.43)
  Change at Week 8: number analyzed (Participants) | 30 | 30 | 27 | 31 | 28 | 36 | 25 | 29 | 28
  Change at Week 8 | -1.6 (0.39) | -1.9 (0.39) | -0.9 (0.41) | -2.1 (0.39) | -2.3 (0.40) | -1.3 (0.42) | -2.4 (0.50) | -2.3 (0.48) | -2.5 (0.48)
  Change at Week 10: number analyzed (Participants) | 29 | 30 | 25 | 29 | 28 | 33 | 24 | 28 | 26
  Change at Week 10 | -1.6 (0.41) | -2.1 (0.40) | -1.6 (0.42) | -2.3 (0.40) | -2.4 (0.41) | -1.1 (0.46) | -2.4 (0.55) | -2.4 (0.53) | -2.4 (0.53)
  Change at Week 12: number analyzed (Participants) | 29 | 29 | 26 | 29 | 28 | 34 | 24 | 29 | 28
  Change at Week 12 | -1.4 (0.49) | -2.1 (0.48) | -1.2 (0.51) | -2.2 (0.48) | -2.4 (0.49) | -0.9 (0.51) | -2.5 (0.62) | -2.5 (0.59) | -2.3 (0.59)
Statistical Analysis 1: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 1: Mixed-effect model with repeated measures (MMRM) analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.8038, MMRM; LS mean difference = 0.3, 90% CI 2-sided [-0.25 to 0.79], Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 1: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.8267, MMRM; LS mean difference = 0.3, 90% CI 2-sided [-0.22 to 0.81], Standard Error of Mean 0.31
Statistical Analysis 3: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.6039, MMRM; LS mean difference = 0.1, 90% CI 2-sided [-0.43 to 0.60], Standard Error of Mean 0.31
Statistical Analysis 4: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.6339, MMRM; LS mean difference = 0.1, 90% CI 2-sided [-0.41 to 0.62], Standard Error of Mean 0.31
Statistical Analysis 5: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.2666, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-0.68 to 0.31], Standard Error of Mean 0.30
Statistical Analysis 6: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.2257, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-0.70 to 0.26], Standard Error of Mean 0.29
Statistical Analysis 7: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.1306, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-0.81 to 0.15], Standard Error of Mean 0.29
Statistical Analysis 8: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 2: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.9704, MMRM; LS mean difference = 0.7, 90% CI 2-sided [0.09 to 1.31], Standard Error of Mean 0.37
Statistical Analysis 9: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 4, analysis 8]; Test type: Superiority; p = 0.8890, MMRM; LS mean difference = 0.5, 90% CI 2-sided [-0.16 to 1.09], Standard Error of Mean 0.38
Statistical Analysis 10: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 4, analysis 8]; Test type: Superiority; p = 0.4506, MMRM; LS mean difference = 0.0, 90% CI 2-sided [-0.66 to 0.57], Standard Error of Mean 0.37
Statistical Analysis 11: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 4, analysis 8]; Test type: Superiority; p = 0.5840, MMRM; LS mean difference = 0.1, 90% CI 2-sided [-0.53 to 0.69], Standard Error of Mean 0.37
Statistical Analysis 12: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 4, analysis 8]; Test type: Superiority; p = 0.0769, MMRM; LS mean difference = -0.5, 90% CI 2-sided [-1.17 to 0.08], Standard Error of Mean 0.38
Statistical Analysis 13: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 4, analysis 8]; Test type: Superiority; p = 0.0242, MMRM; LS mean difference = -0.8, 90% CI 2-sided [-1.39 to -0.13], Standard Error of Mean 0.38
Statistical Analysis 14: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 4, analysis 8]; Test type: Superiority; p = 0.0127, MMRM; LS mean difference = -0.9, 90% CI 2-sided [-1.49 to -0.23], Standard Error of Mean 0.38
Statistical Analysis 15: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 4: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.6693, MMRM; LS mean difference = 0.2, 90% CI 2-sided [-0.54 to 0.93], Standard Error of Mean 0.44
Statistical Analysis 16: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.6742, MMRM; LS mean difference = 0.2, 90% CI 2-sided [-0.55 to 0.96], Standard Error of Mean 0.45
Statistical Analysis 17: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.4486, MMRM; LS mean difference = -0.1, 90% CI 2-sided [-0.79 to 0.67], Standard Error of Mean 0.44
Statistical Analysis 18: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.3219, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-0.93 to 0.53], Standard Error of Mean 0.44
Statistical Analysis 19: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.0096, MMRM; LS mean difference = -1.3, 90% CI 2-sided [-2.21 to -0.39], Standard Error of Mean 0.55
Statistical Analysis 20: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.0862, MMRM; LS mean difference = -0.7, 90% CI 2-sided [-1.64 to 0.15], Standard Error of Mean 0.54
Statistical Analysis 21: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.0111, MMRM; LS mean difference = -1.3, 90% CI 2-sided [-2.15 to -0.36], Standard Error of Mean 0.54
Statistical Analysis 22: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 6: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.6107, MMRM; LS mean difference = 0.1, 90% CI 2-sided [-0.68 to 0.97], Standard Error of Mean 0.50
Statistical Analysis 23: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 4, analysis 22]; Test type: Superiority; p = 0.7240, MMRM; LS mean difference = 0.3, 90% CI 2-sided [-0.54 to 1.15], Standard Error of Mean 0.51
Statistical Analysis 24: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 4, analysis 22]; Test type: Superiority; p = 0.4300, MMRM; LS mean difference = -0.1, 90% CI 2-sided [-0.91 to 0.74], Standard Error of Mean 0.50
Statistical Analysis 25: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 4, analysis 22]; Test type: Superiority; p = 0.0501, MMRM; LS mean difference = -0.8, 90% CI 2-sided [-1.66 to 0.00], Standard Error of Mean 0.50
Statistical Analysis 26: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 4, analysis 22]; Test type: Superiority; p = 0.0157, MMRM; LS mean difference = -1.3, 90% CI 2-sided [-2.23 to -0.30], Standard Error of Mean 0.58
Statistical Analysis 27: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 4, analysis 22]; Test type: Superiority; p = 0.0645, MMRM; LS mean difference = -0.9, 90% CI 2-sided [-1.83 to 0.07], Standard Error of Mean 0.57
Statistical Analysis 28: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 4, analysis 22]; Test type: Superiority; p = 0.0621, MMRM; LS mean difference = -0.9, 90% CI 2-sided [-1.84 to 0.06], Standard Error of Mean 0.57
Statistical Analysis 29: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 8: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.2959, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-1.21 to 0.62], Standard Error of Mean 0.55
Statistical Analysis 30: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 4, analysis 29]; Test type: Superiority; p = 0.9043, MMRM; LS mean difference = 0.7, 90% CI 2-sided [-0.19 to 1.69], Standard Error of Mean 0.57
Statistical Analysis 31: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 4, analysis 29]; Test type: Superiority; p = 0.2014, MMRM; LS mean difference = -0.5, 90% CI 2-sided [-1.38 to 0.45], Standard Error of Mean 0.55
Statistical Analysis 32: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 4, analysis 29]; Test type: Superiority; p = 0.0948, MMRM; LS mean difference = -0.7, 90% CI 2-sided [-1.66 to 0.19], Standard Error of Mean 0.56
Statistical Analysis 33: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 4, analysis 29]; Test type: Superiority; p = 0.0416, MMRM; LS mean difference = -1.1, 90% CI 2-sided [-2.21 to -0.06], Standard Error of Mean 0.65
Statistical Analysis 34: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 4, analysis 29]; Test type: Superiority; p = 0.0454, MMRM; LS mean difference = -1.1, 90% CI 2-sided [-2.14 to -0.03], Standard Error of Mean 0.64
Statistical Analysis 35: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 4, analysis 29]; Test type: Superiority; p = 0.0256, MMRM; LS mean difference = -1.3, 90% CI 2-sided [-2.31 to -0.20], Standard Error of Mean 0.64
Statistical Analysis 36: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 10: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.2326, MMRM; LS mean difference = -0.4, 90% CI 2-sided [-1.36 to 0.53], Standard Error of Mean 0.57
Statistical Analysis 37: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 4, analysis 36]; Test type: Superiority; p = 0.5141, MMRM; LS mean difference = 0.0, 90% CI 2-sided [-0.95 to 0.99], Standard Error of Mean 0.59
Statistical Analysis 38: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 4, analysis 36]; Test type: Superiority; p = 0.1124, MMRM; LS mean difference = -0.7, 90% CI 2-sided [-1.64 to 0.25], Standard Error of Mean 0.57
Statistical Analysis 39: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 4, analysis 36]; Test type: Superiority; p = 0.0983, MMRM; LS mean difference = -0.7, 90% CI 2-sided [-1.70 to 0.21], Standard Error of Mean 0.58
Statistical Analysis 40: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 4, analysis 36]; Test type: Superiority; p = 0.0412, MMRM; LS mean difference = -1.3, 90% CI 2-sided [-2.46 to -0.07], Standard Error of Mean 0.72
Statistical Analysis 41: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 4, analysis 36]; Test type: Superiority; p = 0.0340, MMRM; LS mean difference = -1.3, 90% CI 2-sided [-2.47 to -0.13], Standard Error of Mean 0.71
Statistical Analysis 42: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 4, analysis 36]; Test type: Superiority; p = 0.0379, MMRM; LS mean difference = -1.3, 90% CI 2-sided [-2.44 to -0.09], Standard Error of Mean 0.71
Statistical Analysis 43: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 12: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.1291, MMRM; LS mean difference = -0.8, 90% CI 2-sided [-1.91 to 0.36], Standard Error of Mean 0.68
Statistical Analysis 44: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 4, analysis 43]; Test type: Superiority; p = 0.5776, MMRM; LS mean difference = 0.1, 90% CI 2-sided [-1.03 to 1.30], Standard Error of Mean 0.70
Statistical Analysis 45: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 4, analysis 43]; Test type: Superiority; p = 0.1044, MMRM; LS mean difference = -0.9, 90% CI 2-sided [-2.00 to 0.27], Standard Error of Mean 0.69
Statistical Analysis 46: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 4, analysis 43]; Test type: Superiority; p = 0.0608, MMRM; LS mean difference = -1.1, 90% CI 2-sided [-2.23 to 0.07], Standard Error of Mean 0.69
Statistical Analysis 47: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 4, analysis 43]; Test type: Superiority; p = 0.0309, MMRM; LS mean difference = -1.5, 90% CI 2-sided [-2.84 to -0.18], Standard Error of Mean 0.80
Statistical Analysis 48: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 4, analysis 43]; Test type: Superiority; p = 0.0242, MMRM; LS mean difference = -1.6, 90% CI 2-sided [-2.85 to -0.26], Standard Error of Mean 0.78
Statistical Analysis 49: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 4, analysis 43]; Test type: Superiority; p = 0.0394, MMRM; LS mean difference = -1.4, 90% CI 2-sided [-2.69 to -0.09], Standard Error of Mean 0.78

5. Secondary Outcome: Change From Baseline in PASI Scores at Week 14 and 16
Description: as for outcome 3
Time Frame: Baseline, Week 14 and 16
Population: EAS included all randomized participants who receive at least 1 dose of investigational product (PF-06700841 or placebo) and Week 12 visits were not missing due to COVID-19 pandemic. Here, "number analyzed" signifies the number of participants evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 36 | 37 | 37 | 36 | 37 | 49 | 36 | 35 | 38
Unit on a scale
  Baseline | 6.12 (2.870) | 7.19 (3.370) | 6.46 (2.932) | 6.63 (3.468) | 6.83 (3.137) | 6.08 (2.558) | 7.07 (3.579) | 5.80 (2.765) | 7.94 (4.071)
  Change at Week 14: number analyzed (Participants) | 29 | 26 | 23 | 28 | 28 | 29 | 23 | 25 | 27
  Change at Week 14 | -0.83 (2.379) | -2.24 (2.945) | -0.72 (4.107) | -1.81 (3.228) | -1.87 (2.942) | -0.82 (3.581) | -1.04 (3.732) | -2.06 (3.343) | -1.19 (3.323)
  Change at Week 16: number analyzed (Participants) | 29 | 27 | 23 | 28 | 26 | 31 | 23 | 24 | 26
  Change at Week 16 | -0.46 (2.603) | -2.06 (3.252) | -0.78 (4.223) | -2.10 (3.666) | -1.68 (3.255) | -0.67 (4.008) | -0.71 (3.455) | -1.75 (3.887) | -1.03 (3.351)

6. Secondary Outcome: Percent Change From Baseline in PASI Scores at Week 1, 2, 4, 6, 8, 10 and 12
Description: as for outcome 3
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 32 | 36 | 34 | 35 | 35 | 45 | 35 | 34 | 37
Percent change
  Change at Week 1: number analyzed (Participants) | 32 | 33 | 34 | 35 | 35 | 45 | 32 | 34 | 37
  Change at Week 1 | -15.5 (3.62) | -12.9 (3.57) | -8.2 (3.56) | -10.4 (3.49) | -13.0 (3.51) | -7.4 (3.10) | -9.0 (3.64) | -13.7 (3.58) | -13.5 (3.52)
  Change at Week 2: number analyzed (Participants) | 32 | 36 | 31 | 35 | 35 | 45 | 35 | 32 | 35
  Change at Week 2 | -21.6 (4.25) | -12.4 (4.10) | -12.6 (4.34) | -17.9 (4.13) | -19.8 (4.14) | -11.7 (3.99) | -20.7 (4.60) | -23.3 (4.68) | -24.7 (4.58)
  Change at Week 4: number analyzed (Participants) | 32 | 32 | 28 | 34 | 34 | 45 | 30 | 33 | 33
  Change at Week 4 | -24.1 (4.69) | -20.5 (4.65) | -15.6 (4.90) | -17.6 (4.59) | -25.1 (4.61) | -13.2 (5.69) | -33.9 (6.85) | -24.1 (6.66) | -29.2 (6.64)
  Change at Week 6: number analyzed (Participants) | 31 | 31 | 27 | 31 | 29 | 36 | 28 | 28 | 29
  Change at Week 6 | -23.7 (5.88) | -20.3 (5.83) | -18.4 (6.18) | -21.8 (5.83) | -36.0 (5.92) | -17.8 (6.10) | -36.6 (7.31) | -31.2 (7.12) | -27.5 (7.08)
  Change at Week 8: number analyzed (Participants) | 30 | 30 | 27 | 31 | 28 | 36 | 25 | 29 | 28
  Change at Week 8 | -25.3 (6.48) | -25.6 (6.44) | -14.3 (6.78) | -30.5 (6.41) | -35.9 (6.57) | -18.1 (6.70) | -35.2 (8.07) | -32.4 (7.76) | -34.3 (7.76)
  Change at Week 10: number analyzed (Participants) | 29 | 30 | 25 | 29 | 28 | 33 | 24 | 28 | 26
  Change at Week 10 | -26.8 (6.42) | -27.6 (6.34) | -22.9 (6.73) | -35.3 (6.36) | -36.1 (6.48) | -12.5 (7.62) | -33.4 (9.12) | -35.1 (8.75) | -34.6 (8.77)
  Change at Week 12: number analyzed (Participants) | 29 | 29 | 26 | 29 | 28 | 34 | 24 | 29 | 28
  Change at Week 12 | -20.0 (7.36) | -29.1 (7.30) | -18.5 (7.70) | -33.7 (7.30) | -39.0 (7.47) | -9.6 (8.61) | -34.1 (10.35) | -35.7 (9.84) | -33.7 (9.88)
Statistical Analysis 1: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 1: MMRM analysis contains treatment, visit, and treatment by visit interaction as fixed factors; and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.6917, MMRM; LS mean difference = 2.6, 90% CI 2-sided [-5.86 to 10.97], Standard Error of Mean 5.09
Statistical Analysis 2: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.9241, MMRM; LS mean difference = 7.3, 90% CI 2-sided [-1.09 to 15.69], Standard Error of Mean 5.07
Statistical Analysis 3: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.8443, MMRM; LS mean difference = 5.1, 90% CI 2-sided [-3.21 to 13.42], Standard Error of Mean 5.03
Statistical Analysis 4: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.6911, MMRM; LS mean difference = 2.5, 90% CI 2-sided [-5.82 to 10.86], Standard Error of Mean 5.04
Statistical Analysis 5: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.3676, MMRM; LS mean difference = -1.6, 90% CI 2-sided [-9.56 to 6.31], Standard Error of Mean 4.79
Statistical Analysis 6: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 1: Week 1: MMRM analysis contains treatment, visit, and treatment by visit interaction as fixed factors; and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.0915, MMRM; LS mean difference = -6.3, 90% CI 2-sided [-14.13 to 1.50], Standard Error of Mean 4.72
Statistical Analysis 7: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.0970, MMRM; LS mean difference = -6.2, 90% CI 2-sided [-13.96 to 1.65], Standard Error of Mean 4.72
Statistical Analysis 8: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 2: MMRM analysis contains treatment, visit, and treatment by visit interaction as fixed factors; and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.9389, MMRM; LS mean difference = 9.2, 90% CI 2-sided [-0.59 to 18.97], Standard Error of Mean 5.91
Statistical Analysis 9: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 6, analysis 8]; Test type: Superiority; p = 0.9295, MMRM; LS mean difference = 9.0, 90% CI 2-sided [-1.06 to 19.02], Standard Error of Mean 6.07
Statistical Analysis 10: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 6, analysis 8]; Test type: Superiority; p = 0.7308, MMRM; LS mean difference = 3.7, 90% CI 2-sided [-6.15 to 13.45], Standard Error of Mean 5.92
Statistical Analysis 11: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 6, analysis 8]; Test type: Superiority; p = 0.6199, MMRM; LS mean difference = 1.8, 90% CI 2-sided [-8.01 to 11.64], Standard Error of Mean 5.94
Statistical Analysis 12: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 6, analysis 8]; Test type: Superiority; p = 0.0699, MMRM; LS mean difference = -9.0, 90% CI 2-sided [-19.13 to 1.04], Standard Error of Mean 6.09
Statistical Analysis 13: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 6, analysis 8]; Test type: Superiority; p = 0.0300, MMRM; LS mean difference = -11.6, 90% CI 2-sided [-21.79 to -1.48], Standard Error of Mean 6.14
Statistical Analysis 14: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 6, analysis 8]; Test type: Superiority; p = 0.0168, MMRM; LS mean difference = -13.1, 90% CI 2-sided [-23.15 to -2.98], Standard Error of Mean 6.09
Statistical Analysis 15: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 4: MMRM analysis contains treatment, visit, and treatment by visit interaction as fixed factors; and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.7083, MMRM; LS mean difference = 3.6, 90% CI 2-sided [-7.30 to 14.57], Standard Error of Mean 6.61
Statistical Analysis 16: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p = 0.8955, MMRM; LS mean difference = 8.5, 90% CI 2-sided [-2.66 to 19.75], Standard Error of Mean 6.77
Statistical Analysis 17: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p = 0.8386, MMRM; LS mean difference = 6.5, 90% CI 2-sided [-4.35 to 17.37], Standard Error of Mean 6.56
Statistical Analysis 18: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p = 0.4371, MMRM; LS mean difference = -1.0, 90% CI 2-sided [-11.93 to 9.84], Standard Error of Mean 6.58
Statistical Analysis 19: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p = 0.0108, MMRM; LS mean difference = -20.7, 90% CI 2-sided [-35.42 to -5.92], Standard Error of Mean 8.91
Statistical Analysis 20: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p = 0.1066, MMRM; LS mean difference = -10.9, 90% CI 2-sided [-25.43 to 3.55], Standard Error of Mean 8.75
Statistical Analysis 21: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 6, analysis 15]; Test type: Superiority; p = 0.0344, MMRM; LS mean difference = -16.0, 90% CI 2-sided [-30.54 to -1.55], Standard Error of Mean 8.76
Statistical Analysis 22: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 6: MMRM analysis contains treatment, visit, and treatment by visit interaction as fixed factors; and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.6594, MMRM; LS mean difference = 3.4, 90% CI 2-sided [-10.30 to 17.13], Standard Error of Mean 8.29
Statistical Analysis 23: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 6, analysis 22]; Test type: Superiority; p = 0.7307, MMRM; LS mean difference = 5.3, 90% CI 2-sided [-8.85 to 19.36], Standard Error of Mean 8.52
Statistical Analysis 24: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 6, analysis 22]; Test type: Superiority; p = 0.5914, MMRM; LS mean difference = 1.9, 90% CI 2-sided [-11.78 to 15.61], Standard Error of Mean 8.28
Statistical Analysis 25: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 6, analysis 22]; Test type: Superiority; p = 0.0709, MMRM; LS mean difference = -12.3, 90% CI 2-sided [-26.13 to 1.49], Standard Error of Mean 8.34
Statistical Analysis 26: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 6, analysis 22]; Test type: Superiority; p = 0.0253, MMRM; LS mean difference = -18.8, 90% CI 2-sided [-34.55 to -3.01], Standard Error of Mean 9.53
Statistical Analysis 27: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 6, analysis 22]; Test type: Superiority; p = 0.0780, MMRM; LS mean difference = -13.4, 90% CI 2-sided [-28.89 to 2.15], Standard Error of Mean 9.38
Statistical Analysis 28: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 6, analysis 22]; Test type: Superiority; p = 0.1516, MMRM; LS mean difference = -9.7, 90% CI 2-sided [-25.17 to 5.83], Standard Error of Mean 9.36
Statistical Analysis 29: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 8: MMRM analysis contains treatment, visit, and treatment by visit interaction as fixed factors; and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.4861, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-15.45 to 14.81], Standard Error of Mean 9.14
Statistical Analysis 30: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 6, analysis 29]; Test type: Superiority; p = 0.8795, MMRM; LS mean difference = 11.0, 90% CI 2-sided [-4.48 to 26.55], Standard Error of Mean 9.38
Statistical Analysis 31: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 6, analysis 29]; Test type: Superiority; p = 0.2867, MMRM; LS mean difference = -5.1, 90% CI 2-sided [-20.22 to 9.94], Standard Error of Mean 9.11
Statistical Analysis 32: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 6, analysis 29]; Test type: Superiority; p = 0.1267, MMRM; LS mean difference = -10.6, 90% CI 2-sided [-25.86 to 4.69], Standard Error of Mean 9.23
Statistical Analysis 33: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 6, analysis 29]; Test type: Superiority; p = 0.0526, MMRM; LS mean difference = -17.1, 90% CI 2-sided [-34.48 to 0.26], Standard Error of Mean 10.49
Statistical Analysis 34: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 6, analysis 29]; Test type: Superiority; p = 0.0827, MMRM; LS mean difference = -14.3, 90% CI 2-sided [-31.26 to 2.68], Standard Error of Mean 10.25
Statistical Analysis 35: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 6, analysis 29]; Test type: Superiority; p = 0.0592, MMRM; LS mean difference = -16.1, 90% CI 2-sided [-33.12 to 0.86], Standard Error of Mean 10.26
Statistical Analysis 36: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 10: MMRM analysis contains treatment, visit, and treatment by visit interaction as fixed factors; and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.4657, MMRM; LS mean difference = -0.8, 90% CI 2-sided [-15.72 to 14.16], Standard Error of Mean 9.03
Statistical Analysis 37: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 6, analysis 36]; Test type: Superiority; p = 0.6612, MMRM; LS mean difference = 3.9, 90% CI 2-sided [-11.52 to 19.26], Standard Error of Mean 9.30
Statistical Analysis 38: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 6, analysis 36]; Test type: Superiority; p = 0.1749, MMRM; LS mean difference = -8.5, 90% CI 2-sided [-23.42 to 6.48], Standard Error of Mean 9.03
Statistical Analysis 39: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 6, analysis 36]; Test type: Superiority; p = 0.1548, MMRM; LS mean difference = -9.3, 90% CI 2-sided [-24.39 to 5.80], Standard Error of Mean 9.12
Statistical Analysis 40: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 6, analysis 36]; Test type: Superiority; p = 0.0400, MMRM; LS mean difference = -21.0, 90% CI 2-sided [-40.67 to -1.28], Standard Error of Mean 11.89
Statistical Analysis 41: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 6, analysis 36]; Test type: Superiority; p = 0.0267, MMRM; LS mean difference = -22.6, 90% CI 2-sided [-41.82 to -3.39], Standard Error of Mean 11.60
Statistical Analysis 42: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 6, analysis 36]; Test type: Superiority; p = 0.0295, MMRM; LS mean difference = -22.2, 90% CI 2-sided [-41.42 to -2.89], Standard Error of Mean 11.63
Statistical Analysis 43: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 12: MMRM analysis contains treatment, visit, and treatment by visit interaction as fixed factors; and baseline value as a covariate. Unstructured covariance matrix was used for model errors; Test type: Superiority; p = 0.1903, MMRM; LS mean difference = -9.1, 90% CI 2-sided [-26.30 to 8.05], Standard Error of Mean 10.38
Statistical Analysis 44: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 6, analysis 43]; Test type: Superiority; p = 0.5530, MMRM; LS mean difference = 1.4, 90% CI 2-sided [-16.21 to 19.06], Standard Error of Mean 10.65
Statistical Analysis 45: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 6, analysis 43]; Test type: Superiority; p = 0.0933, MMRM; LS mean difference = -13.8, 90% CI 2-sided [-30.92 to 3.40], Standard Error of Mean 10.37
Statistical Analysis 46: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 6, analysis 43]; Test type: Superiority; p = 0.0360, MMRM; LS mean difference = -19.0, 90% CI 2-sided [-36.37 to -1.65], Standard Error of Mean 10.49
Statistical Analysis 47: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 6, analysis 43]; Test type: Superiority; p = 0.0354, MMRM; LS mean difference = -24.5, 90% CI 2-sided [-46.85 to -2.23], Standard Error of Mean 13.46
Statistical Analysis 48: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 6, analysis 43]; Test type: Superiority; p = 0.0239, MMRM; LS mean difference = -26.1, 90% CI 2-sided [-47.77 to -4.46], Standard Error of Mean 13.07
Statistical Analysis 49: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 6, analysis 43]; Test type: Superiority; p = 0.0342, MMRM; LS mean difference = -24.1, 90% CI 2-sided [-45.84 to -2.38], Standard Error of Mean 13.11

7. Secondary Outcome: Percent Change From Baseline in PASI Scores at Week 14 and 16
Description: as for outcome 3
Time Frame: Baseline, Week 14 and 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 36 | 37 | 37 | 36 | 37 | 49 | 36 | 35 | 38
Percent change
  Baseline | 6.12 (2.870) | 7.19 (3.370) | 6.46 (2.932) | 6.63 (3.468) | 6.83 (3.137) | 6.08 (2.558) | 7.07 (3.579) | 5.80 (2.765) | 7.94 (4.071)
  Change at Week 14: number analyzed (Participants) | 29 | 26 | 23 | 28 | 28 | 29 | 23 | 25 | 27
  Change at Week 14 | -12.76 (49.660) | -25.94 (40.339) | -8.58 (59.407) | -23.14 (47.501) | -30.07 (40.222) | -5.74 (74.846) | -14.18 (58.599) | -27.56 (45.370) | -19.74 (49.727)
  Change at Week 16: number analyzed (Participants) | 29 | 27 | 23 | 28 | 26 | 31 | 23 | 24 | 26
  Change at Week 16 | -4.72 (56.401) | -23.01 (44.766) | -9.00 (60.088) | -29.24 (52.608) | -27.17 (41.153) | -3.75 (83.415) | -9.99 (60.306) | -24.09 (48.685) | -21.12 (52.521)

8. Secondary Outcome: Absolute Peak-Pruritus Numerical Rating Scale (PP-NRS) Score at Baseline, Week 1, 2, 4, 6, 8, 10 and 12
Description: Participants were asked to assess their itch intensity over the past 24 hours, on a scale from 0 (no itching) to 10 (worst possible itching). Higher scores indicated worse itch.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 35 | 36 | 34 | 36 | 36 | 48 | 35 | 35 | 31
Unit on a scale
  Baseline: number analyzed (Participants) | 33 | 34 | 33 | 29 | 36 | 43 | 33 | 32 | 30
  Baseline | 4.6 (0.31) | 4.4 (0.30) | 4.5 (0.31) | 4.1 (0.33) | 4.5 (0.29) | 4.9 (0.28) | 4.8 (0.32) | 4.4 (0.32) | 5.4 (0.34)
  Week 1: number analyzed (Participants) | 35 | 36 | 34 | 36 | 36 | 47 | 34 | 34 | 29
  Week 1 | 4.1 (0.31) | 3.9 (0.30) | 3.6 (0.31) | 3.5 (0.33) | 3.6 (0.30) | 4.0 (0.28) | 3.8 (0.32) | 3.4 (0.32) | 3.7 (0.35)
  Week 2: number analyzed (Participants) | 35 | 36 | 33 | 35 | 35 | 48 | 35 | 35 | 31
  Week 2 | 3.6 (0.31) | 3.5 (0.31) | 3.3 (0.31) | 3.2 (0.33) | 3.5 (0.30) | 3.5 (0.28) | 3.6 (0.32) | 2.9 (0.32) | 3.4 (0.35)
  Week 4: number analyzed (Participants) | 31 | 31 | 27 | 33 | 34 | 45 | 29 | 31 | 31
  Week 4 | 3.5 (0.32) | 3.7 (0.32) | 3.2 (0.33) | 3.2 (0.34) | 3.2 (0.30) | 3.4 (0.29) | 3.0 (0.34) | 3.0 (0.34) | 3.4 (0.36)
  Week 6: number analyzed (Participants) | 32 | 30 | 25 | 31 | 28 | 38 | 27 | 27 | 27
  Week 6 | 3.5 (0.32) | 4.0 (0.32) | 3.5 (0.34) | 3.2 (0.34) | 2.9 (0.32) | 3.6 (0.31) | 2.8 (0.35) | 3.0 (0.35) | 2.9 (0.38)
  Week 8: number analyzed (Participants) | 30 | 31 | 26 | 31 | 26 | 36 | 24 | 27 | 27
  Week 8 | 3.1 (0.32) | 3.4 (0.32) | 3.2 (0.33) | 3.1 (0.34) | 2.8 (0.32) | 3.3 (0.32) | 2.7 (0.37) | 2.9 (0.35) | 2.7 (0.38)
  Week 10: number analyzed (Participants) | 29 | 28 | 25 | 29 | 28 | 31 | 24 | 28 | 24
  Week 10 | 3.3 (0.33) | 3.0 (0.33) | 3.0 (0.34) | 3.1 (0.35) | 2.3 (0.32) | 4.1 (0.33) | 2.8 (0.36) | 2.9 (0.35) | 3.6 (0.39)
  Week 12: number analyzed (Participants) | 29 | 29 | 26 | 29 | 27 | 31 | 23 | 28 | 25
  Week 12 | 3.4 (0.33) | 3.1 (0.33) | 3.1 (0.33) | 3.0 (0.35) | 2.6 (0.32) | 4.0 (0.32) | 2.7 (0.37) | 3.0 (0.35) | 3.2 (0.40)
Statistical Analysis 1: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Baseline: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Compound symmetry covariance matrix was used for model errors; Test type: Superiority; p = 0.3279, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-0.91 to 0.52], Standard Error of Mean 0.43
Statistical Analysis 2: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.3566, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-0.88 to 0.56], Standard Error of Mean 0.44
Statistical Analysis 3: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.1165, MMRM; LS mean difference = -0.5, 90% CI 2-sided [-1.29 to 0.21], Standard Error of Mean 0.45
Statistical Analysis 4: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.3633, MMRM; LS mean difference = -0.1, 90% CI 2-sided [-0.85 to 0.55], Standard Error of Mean 0.43
Statistical Analysis 5: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.3766, MMRM; LS mean difference = -0.1, 90% CI 2-sided [-0.83 to 0.56], Standard Error of Mean 0.42
Statistical Analysis 6: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.1179, MMRM; LS mean difference = -0.5, 90% CI 2-sided [-1.22 to 0.20], Standard Error of Mean 0.43
Statistical Analysis 7: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.8647, MMRM; LS mean difference = 0.5, 90% CI 2-sided [-0.24 to 1.20], Standard Error of Mean 0.44
Statistical Analysis 8: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 1: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Compound symmetry covariance matrix was used for model errors; Test type: Superiority; p = 0.3294, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-0.90 to 0.52], Standard Error of Mean 0.43
Statistical Analysis 9: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 8, analysis 8]; Test type: Superiority; p = 0.1231, MMRM; LS mean difference = -0.5, 90% CI 2-sided [-1.23 to 0.21], Standard Error of Mean 0.44
Statistical Analysis 10: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 8, analysis 8]; Test type: Superiority; p = 0.0878, MMRM; LS mean difference = -0.6, 90% CI 2-sided [-1.37 to 0.13], Standard Error of Mean 0.45
Statistical Analysis 11: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 8, analysis 8]; Test type: Superiority; p = 0.1225, MMRM; LS mean difference = -0.5, 90% CI 2-sided [-1.20 to 0.21], Standard Error of Mean 0.43
Statistical Analysis 12: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 8, analysis 8]; Test type: Superiority; p = 0.3663, MMRM; LS mean difference = -0.1, 90% CI 2-sided [-0.85 to 0.56], Standard Error of Mean 0.43
Statistical Analysis 13: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 8, analysis 8]; Test type: Superiority; p = 0.0929, MMRM; LS mean difference = -0.6, 90% CI 2-sided [-1.27 to 0.14], Standard Error of Mean 0.43
Statistical Analysis 14: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 8, analysis 8]; Test type: Superiority; p = 0.3111, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-0.95 to 0.51], Standard Error of Mean 0.44
Statistical Analysis 15: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 2: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Compound symmetry covariance matrix was used for model errors; Test type: Superiority; p = 0.4745, MMRM; LS mean difference = 0.0, 90% CI 2-sided [-0.74 to 0.69], Standard Error of Mean 0.43
Statistical Analysis 16: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 8, analysis 15]; Test type: Superiority; p = 0.2409, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-1.03 to 0.42], Standard Error of Mean 0.44
Statistical Analysis 17: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 8, analysis 15]; Test type: Superiority; p = 0.2018, MMRM; LS mean difference = -0.4, 90% CI 2-sided [-1.13 to 0.37], Standard Error of Mean 0.45
Statistical Analysis 18: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 8, analysis 15]; Test type: Superiority; p = 0.3925, MMRM; LS mean difference = -0.1, 90% CI 2-sided [-0.83 to 0.59], Standard Error of Mean 0.43
Statistical Analysis 19: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 8, analysis 15]; Test type: Superiority; p = 0.5348, MMRM; LS mean difference = 0.0, 90% CI 2-sided [-0.66 to 0.73], Standard Error of Mean 0.42
Statistical Analysis 20: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 8, analysis 15]; Test type: Superiority; p = 0.0739, MMRM; LS mean difference = -0.6, 90% CI 2-sided [-1.33 to 0.09], Standard Error of Mean 0.43
Statistical Analysis 21: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 8, analysis 15]; Test type: Superiority; p = 0.4014, MMRM; LS mean difference = -0.1, 90% CI 2-sided [-0.84 to 0.62], Standard Error of Mean 0.44
Statistical Analysis 22: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 4: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Compound symmetry covariance matrix was used for model errors; Test type: Superiority; p = 0.6588, MMRM; LS mean difference = 0.2, 90% CI 2-sided [-0.56 to 0.93], Standard Error of Mean 0.45
Statistical Analysis 23: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 8, analysis 22]; Test type: Superiority; p = 0.2997, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-1.00 to 0.52], Standard Error of Mean 0.46
Statistical Analysis 24: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 4:MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Compound symmetry covariance matrix was used for model errors; Test type: Superiority; p = 0.2518, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-1.08 to 0.46], Standard Error of Mean 0.47
Statistical Analysis 25: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 8, analysis 22]; Test type: Superiority; p = 0.2634, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-1.00 to 0.45], Standard Error of Mean 0.44
Statistical Analysis 26: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 8, analysis 22]; Test type: Superiority; p = 0.1999, MMRM; LS mean difference = -0.4, 90% CI 2-sided [-1.11 to 0.36], Standard Error of Mean 0.45
Statistical Analysis 27: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 8, analysis 22]; Test type: Superiority; p = 0.1847, MMRM; LS mean difference = -0.4, 90% CI 2-sided [-1.13 to 0.33], Standard Error of Mean 0.44
Statistical Analysis 28: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 8, analysis 22]; Test type: Superiority; p = 0.4569, MMRM; LS mean difference = 0.0, 90% CI 2-sided [-0.81 to 0.71], Standard Error of Mean 0.46
Statistical Analysis 29: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 6: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Compound symmetry covariance matrix was used for model errors; Test type: Superiority; p = 0.8536, MMRM; LS mean difference = 0.5, 90% CI 2-sided [-0.27 to 1.22], Standard Error of Mean 0.45
Statistical Analysis 30: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 6:MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Compound symmetry covariance matrix was used for model errors; Test type: Superiority; p = 0.4812, MMRM; LS mean difference = 0.0, 90% CI 2-sided [-0.79 to 0.74], Standard Error of Mean 0.46
Statistical Analysis 31: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 8, analysis 29]; Test type: Superiority; p = 0.2276, MMRM; LS mean difference = -0.4, 90% CI 2-sided [-1.13 to 0.42], Standard Error of Mean 0.47
Statistical Analysis 32: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 8, analysis 29]; Test type: Superiority; p = 0.0895, MMRM; LS mean difference = -0.6, 90% CI 2-sided [-1.34 to 0.14], Standard Error of Mean 0.45
Statistical Analysis 33: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 8, analysis 29]; Test type: Superiority; p = 0.0411, MMRM; LS mean difference = -0.8, 90% CI 2-sided [-1.58 to -0.04], Standard Error of Mean 0.47
Statistical Analysis 34: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 8, analysis 29]; Test type: Superiority; p = 0.0928, MMRM; LS mean difference = -0.6, 90% CI 2-sided [-1.40 to 0.15], Standard Error of Mean 0.47
Statistical Analysis 35: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 8, analysis 29]; Test type: Superiority; p = 0.0799, MMRM; LS mean difference = -0.7, 90% CI 2-sided [-1.48 to 0.12], Standard Error of Mean 0.49
Statistical Analysis 36: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 8: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Compound symmetry covariance matrix was used for model errors; Test type: Superiority; p = 0.7872, MMRM; LS mean difference = 0.4, 90% CI 2-sided [-0.39 to 1.11], Standard Error of Mean 0.46
Statistical Analysis 37: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 8, analysis 36]; Test type: Superiority; p = 0.6294, MMRM; LS mean difference = 0.2, 90% CI 2-sided [-0.61 to 0.92], Standard Error of Mean 0.47
Statistical Analysis 38: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 8, analysis 36]; Test type: Superiority; p = 0.5174, MMRM; LS mean difference = 0.0, 90% CI 2-sided [-0.76 to 0.80], Standard Error of Mean 0.48
Statistical Analysis 39: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 8, analysis 36]; Test type: Superiority; p = 0.3136, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-0.98 to 0.53], Standard Error of Mean 0.46
Statistical Analysis 40: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 8, analysis 36]; Test type: Superiority; p = 0.1020, MMRM; LS mean difference = -0.6, 90% CI 2-sided [-1.42 to 0.18], Standard Error of Mean 0.48
Statistical Analysis 41: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 8, analysis 36]; Test type: Superiority; p = 0.1923, MMRM; LS mean difference = -0.4, 90% CI 2-sided [-1.20 to 0.37], Standard Error of Mean 0.47
Statistical Analysis 42: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 8, analysis 36]; Test type: Superiority; p = 0.0997, MMRM; LS mean difference = -0.6, 90% CI 2-sided [-1.44 to 0.18], Standard Error of Mean 0.49
Statistical Analysis 43: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 10: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Compound symmetry covariance matrix was used for model errors; Test type: Superiority; p = 0.2497, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-1.08 to 0.45], Standard Error of Mean 0.47
Statistical Analysis 44: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 8, analysis 43]; Test type: Superiority; p = 0.2568, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-1.08 to 0.47], Standard Error of Mean 0.47
Statistical Analysis 45: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 8, analysis 43]; Test type: Superiority; p = 0.3730, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-0.95 to 0.64], Standard Error of Mean 0.48
Statistical Analysis 46: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 8, analysis 43]; Test type: Superiority; p = 0.0137, MMRM; LS mean difference = -1.0, 90% CI 2-sided [-1.76 to -0.26], Standard Error of Mean 0.46
Statistical Analysis 47: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 8, analysis 43]; Test type: Superiority; p = 0.0055, MMRM; LS mean difference = -1.3, 90% CI 2-sided [-2.06 to -0.44], Standard Error of Mean 0.49
Statistical Analysis 48: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 8, analysis 43]; Test type: Superiority; p = 0.0069, MMRM; LS mean difference = -1.2, 90% CI 2-sided [-1.99 to -0.40], Standard Error of Mean 0.48
Statistical Analysis 49: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 8, analysis 43]; Test type: Superiority; p = 0.1648, MMRM; LS mean difference = -0.5, 90% CI 2-sided [-1.34 to 0.34], Standard Error of Mean 0.51
Statistical Analysis 50: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 12: MMRM analysis contained treatment, visit, and treatment by visit interaction as fixed factors, and baseline value as a covariate. Compound symmetry covariance matrix was used for model errors; Test type: Superiority; p = 0.2931, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-1.02 to 0.51], Standard Error of Mean 0.46
Statistical Analysis 51: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 8, analysis 50]; Test type: Superiority; p = 0.3047, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-1.01 to 0.53], Standard Error of Mean 0.47
Statistical Analysis 52: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 8, analysis 50]; Test type: Superiority; p = 0.1924, MMRM; LS mean difference = -0.4, 90% CI 2-sided [-1.22 to 0.38], Standard Error of Mean 0.48
Statistical Analysis 53: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 8, analysis 50]; Test type: Superiority; p = 0.0465, MMRM; LS mean difference = -0.8, 90% CI 2-sided [-1.52 to -0.02], Standard Error of Mean 0.46
Statistical Analysis 54: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 8, analysis 50]; Test type: Superiority; p = 0.0048, MMRM; LS mean difference = -1.3, 90% CI 2-sided [-2.08 to -0.47], Standard Error of Mean 0.49
Statistical Analysis 55: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 8, analysis 50]; Test type: Superiority; p = 0.0186, MMRM; LS mean difference = -1.0, 90% CI 2-sided [-1.78 to -0.21], Standard Error of Mean 0.48
Statistical Analysis 56: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 8, analysis 50]; Test type: Superiority; p = 0.0675, MMRM; LS mean difference = -0.8, 90% CI 2-sided [-1.61 to 0.08], Standard Error of Mean 0.51

9. Secondary Outcome: Absolute PP-NRS Score at Week 14 and 16
Description: as for outcome 8
Time Frame: Week 14 and 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 28 | 27 | 24 | 24 | 27 | 30 | 23 | 25 | 23
Unit on a scale
  Week 14: number analyzed (Participants) | 28 | 25 | 24 | 24 | 27 | 27 | 23 | 25 | 23
  Week 14 | 5.2 (3.02) | 2.6 (2.52) | 2.8 (2.38) | 2.4 (2.39) | 3.2 (2.38) | 4.0 (2.77) | 3.5 (2.89) | 2.8 (2.57) | 5.5 (2.81)
  Week 16: number analyzed (Participants) | 27 | 27 | 23 | 24 | 25 | 30 | 22 | 22 | 19
  Week 16 | 4.9 (2.93) | 3.2 (2.75) | 3.1 (2.63) | 2.5 (2.45) | 3.2 (2.42) | 3.8 (2.69) | 3.4 (2.77) | 3.5 (2.91) | 5.8 (2.76)

10. Secondary Outcome: Change From Baseline in PP-NRS Score at Week 1, 2, 4, 6, 8, 10 and 12
Description: as for outcome 8
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10 and 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 33 | 34 | 32 | 29 | 35 | 43 | 33 | 32 | 28
Unit on a scale
  Change at Week 1: number analyzed (Participants) | 33 | 34 | 32 | 29 | 35 | 43 | 32 | 32 | 28
  Change at Week 1 | -0.4 (0.23) | -0.6 (0.23) | -0.9 (0.23) | -0.9 (0.25) | -0.9 (0.22) | -0.9 (0.24) | -1.0 (0.27) | -1.4 (0.28) | -1.2 (0.30)
  Change at Week 2: number analyzed (Participants) | 33 | 33 | 31 | 29 | 34 | 43 | 33 | 32 | 28
  Change at Week 2 | -0.9 (0.28) | -0.9 (0.27) | -1.1 (0.28) | -1.2 (0.30) | -1.0 (0.27) | -1.3 (0.25) | -1.3 (0.29) | -1.9 (0.30) | -1.5 (0.32)
  Change at Week 4: number analyzed (Participants) | 29 | 28 | 26 | 27 | 33 | 40 | 27 | 28 | 25
  Change at Week 4 | -1.0 (0.33) | -0.8 (0.33) | -1.0 (0.34) | -1.2 (0.36) | -1.2 (0.32) | -1.3 (0.32) | -1.7 (0.38) | -1.7 (0.38) | -1.6 (0.41)
  Change at Week 6: number analyzed (Participants) | 30 | 28 | 24 | 25 | 28 | 32 | 25 | 25 | 22
  Change at Week 6 | -0.9 (0.36) | -0.4 (0.36) | -1.0 (0.38) | -1.2 (0.39) | -1.6 (0.36) | -1.1 (0.31) | -1.9 (0.36) | -1.8 (0.36) | -2.1 (0.39)
  Change at Week 8: number analyzed (Participants) | 28 | 28 | 25 | 25 | 26 | 30 | 22 | 25 | 22
  Change at Week 8 | -1.4 (0.38) | -1.1 (0.38) | -1.2 (0.39) | -1.3 (0.41) | -1.6 (0.38) | -1.2 (0.38) | -2.2 (0.44) | -1.8 (0.43) | -2.2 (0.46)
  Change at Week 10: number analyzed (Participants) | 27 | 25 | 24 | 23 | 28 | 26 | 23 | 26 | 20
  Change at Week 10 | -1.1 (0.43) | -1.4 (0.44) | -1.3 (0.45) | -1.2 (0.46) | -2.1 (0.42) | -0.5 (0.39) | -2.1 (0.44) | -1.9 (0.42) | -1.2 (0.47)
  Change at Week 12: number analyzed (Participants) | 27 | 26 | 25 | 23 | 27 | 28 | 22 | 26 | 19
  Change at Week 12 | -1.0 (0.42) | -1.3 (0.43) | -1.2 (0.44) | -1.3 (0.45) | -1.8 (0.42) | -0.6 (0.41) | -2.3 (0.47) | -1.8 (0.44) | -1.5 (0.49)
Statistical Analysis 1: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.3232, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-0.69 to 0.39], Standard Error of Mean 0.33
Statistical Analysis 2: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0736, MMRM; LS mean difference = -0.5, 90% CI 2-sided [-1.03 to 0.07], Standard Error of Mean 0.33
Statistical Analysis 3: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0743, MMRM; LS mean difference = -0.5, 90% CI 2-sided [-1.07 to 0.07], Standard Error of Mean 0.35
Statistical Analysis 4: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0641, MMRM; LS mean difference = -0.5, 90% CI 2-sided [-1.03 to 0.04], Standard Error of Mean 0.32
Statistical Analysis 5: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.3887, MMRM; LS mean difference = -0.1, 90% CI 2-sided [-0.71 to 0.50], Standard Error of Mean 0.36
Statistical Analysis 6: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.0767, MMRM; LS mean difference = -0.5, 90% CI 2-sided [-1.15 to 0.08], Standard Error of Mean 0.37
Statistical Analysis 7: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.2529, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-0.89 to 0.38], Standard Error of Mean 0.38
Statistical Analysis 8: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; [analysis description as in outcome 4, analysis 8]; Test type: Superiority; p = 0.5304, MMRM; LS mean difference = 0.0, 90% CI 2-sided [-0.61 to 0.67], Standard Error of Mean 0.39
Statistical Analysis 9: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 4, analysis 8]; Test type: Superiority; p = 0.2920, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-0.87 to 0.43], Standard Error of Mean 0.39
Statistical Analysis 10: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 4, analysis 8]; Test type: Superiority; p = 0.2593, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-0.70 to 0.57], Standard Error of Mean 0.41
Statistical Analysis 11: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 4, analysis 8]; Test type: Superiority; p = 0.4310, MMRM; LS mean difference = -0.1, 90% CI 2-sided [-0.70 to 0.57], Standard Error of Mean 0.38
Statistical Analysis 12: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 4, analysis 8]; Test type: Superiority; p = 0.5477, MMRM; LS mean difference = 0.0, 90% CI 2-sided [-0.59 to 0.69], Standard Error of Mean 0.39
Statistical Analysis 13: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 4, analysis 8]; Test type: Superiority; p = 0.0696, MMRM; LS mean difference = -0.6, 90% CI 2-sided [-1.24 to 0.07], Standard Error of Mean 0.39
Statistical Analysis 14: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 4, analysis 8]; Test type: Superiority; p = 0.3583, MMRM; LS mean difference = -0.1, 90% CI 2-sided [-0.82 to 0.53], Standard Error of Mean 0.41
Statistical Analysis 15: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.6826, MMRM; LS mean difference = 0.2, 90% CI 2-sided [-0.56 to 1.01], Standard Error of Mean 0.47
Statistical Analysis 16: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.4570, MMRM; LS mean difference = -0.1, 90% CI 2-sided [-0.84 to 0.74], Standard Error of Mean 0.48
Statistical Analysis 17: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.3265, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-1.03 to 0.59], Standard Error of Mean 0.49
Statistical Analysis 18: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.3039, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-1.00 to 0.53], Standard Error of Mean 0.46
Statistical Analysis 19: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.2086, MMRM; LS mean difference = -0.4, 90% CI 2-sided [-1.23 to 0.42], Standard Error of Mean 0.50
Statistical Analysis 20: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.2172, MMRM; LS mean difference = -0.4, 90% CI 2-sided [-1.22 to 0.44], Standard Error of Mean 0.50
Statistical Analysis 21: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 4, analysis 15]; Test type: Superiority; p = 0.2855, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-1.16 to 0.57], Standard Error of Mean 0.52
Statistical Analysis 22: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; [analysis description as in outcome 4, analysis 22]; Test type: Superiority; p = 0.8372, MMRM; LS mean difference = 0.5, 90% CI 2-sided [-0.34 to 1.36], Standard Error of Mean 0.51
Statistical Analysis 23: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 4, analysis 22]; Test type: Superiority; p = 0.4792, MMRM; LS mean difference = 0.0, 90% CI 2-sided [-0.89 to 0.84], Standard Error of Mean 0.52
Statistical Analysis 24: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 4, analysis 22]; Test type: Superiority; p = 0.3331, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-1.12 to 0.65], Standard Error of Mean 0.53
Statistical Analysis 25: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 4, analysis 22]; Test type: Superiority; p = 0.1080, MMRM; LS mean difference = -0.6, 90% CI 2-sided [-1.47 to 0.21], Standard Error of Mean 0.51
Statistical Analysis 26: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 4, analysis 22]; Test type: Superiority; p = 0.0455, MMRM; LS mean difference = -0.8, 90% CI 2-sided [-1.61 to -0.02], Standard Error of Mean 0.48
Statistical Analysis 27: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 4, analysis 22]; Test type: Superiority; p = 0.0761, MMRM; LS mean difference = -0.7, 90% CI 2-sided [-1.49 to 0.10], Standard Error of Mean 0.48
Statistical Analysis 28: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 4, analysis 22]; Test type: Superiority; p = 0.0273, MMRM; LS mean difference = -1.0, 90% CI 2-sided [-1.80 to -0.14], Standard Error of Mean 0.50
Statistical Analysis 29: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; [analysis description as in outcome 4, analysis 29]; Test type: Superiority; p = 0.7214, MMRM; LS mean difference = 0.3, 90% CI 2-sided [-0.57 to 1.20], Standard Error of Mean 0.54
Statistical Analysis 30: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 4, analysis 29]; Test type: Superiority; p = 0.6132, MMRM; LS mean difference = 0.2, 90% CI 2-sided [-0.75 to 1.06], Standard Error of Mean 0.55
Statistical Analysis 31: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 4, analysis 29]; Test type: Superiority; p = 0.5704, MMRM; LS mean difference = 0.1, 90% CI 2-sided [-0.83 to 1.02], Standard Error of Mean 0.56
Statistical Analysis 32: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 4, analysis 29]; Test type: Superiority; p = 0.3449, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-1.10 to 0.67], Standard Error of Mean 0.53
Statistical Analysis 33: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 4, analysis 29]; Test type: Superiority; p = 0.0493, MMRM; LS mean difference = -1.0, 90% CI 2-sided [-1.94 to 0.00], Standard Error of Mean 0.58
Statistical Analysis 34: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 4, analysis 29]; Test type: Superiority; p = 0.1490, MMRM; LS mean difference = -0.6, 90% CI 2-sided [-1.55 to 0.35], Standard Error of Mean 0.57
Statistical Analysis 35: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 4, analysis 29]; Test type: Superiority; p = 0.0540, MMRM; LS mean difference = -1.0, 90% CI 2-sided [-1.96 to 0.02], Standard Error of Mean 0.60
Statistical Analysis 36: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; [analysis description as in outcome 4, analysis 36]; Test type: Superiority; p = 0.3119, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-1.32 to 0.71], Standard Error of Mean 0.61
Statistical Analysis 37: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 4, analysis 36]; Test type: Superiority; p = 0.3947, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-1.20 to 0.86], Standard Error of Mean 0.62
Statistical Analysis 38: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 4, analysis 36]; Test type: Superiority; p = 0.4205, MMRM; LS mean difference = -0.1, 90% CI 2-sided [-1.18 to 0.93], Standard Error of Mean 0.64
Statistical Analysis 39: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 4, analysis 36]; Test type: Superiority; p = 0.0472, MMRM; LS mean difference = -1.0, 90% CI 2-sided [-2.02 to -0.02], Standard Error of Mean 0.60
Statistical Analysis 40: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 4, analysis 36]; Test type: Superiority; p = 0.0044, MMRM; LS mean difference = -1.6, 90% CI 2-sided [-2.55 to -0.60], Standard Error of Mean 0.59
Statistical Analysis 41: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 4, analysis 36]; Test type: Superiority; p = 0.0098, MMRM; LS mean difference = -1.4, 90% CI 2-sided [-2.32 to -0.41], Standard Error of Mean 0.58
Statistical Analysis 42: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 4, analysis 36]; Test type: Superiority; p = 0.1285, MMRM; LS mean difference = -0.7, 90% CI 2-sided [-1.71 to 0.32], Standard Error of Mean 0.61
Statistical Analysis 43: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; [analysis description as in outcome 4, analysis 43]; Test type: Superiority; p = 0.3243, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-1.27 to 0.72], Standard Error of Mean 0.60
Statistical Analysis 44: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; [analysis description as in outcome 4, analysis 43]; Test type: Superiority; p = 0.3795, MMRM; LS mean difference = -0.2, 90% CI 2-sided [-1.20 to 0.82], Standard Error of Mean 0.61
Statistical Analysis 45: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; [analysis description as in outcome 4, analysis 43]; Test type: Superiority; p = 0.3070, MMRM; LS mean difference = -0.3, 90% CI 2-sided [-1.35 to 0.72], Standard Error of Mean 0.62
Statistical Analysis 46: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; [analysis description as in outcome 4, analysis 43]; Test type: Superiority; p = 0.1014, MMRM; LS mean difference = -0.8, 90% CI 2-sided [-1.74 to 0.22], Standard Error of Mean 0.59
Statistical Analysis 47: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; [analysis description as in outcome 4, analysis 43]; Test type: Superiority; p = 0.0033, MMRM; LS mean difference = -1.7, 90% CI 2-sided [-2.75 to -0.69], Standard Error of Mean 0.62
Statistical Analysis 48: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; [analysis description as in outcome 4, analysis 43]; Test type: Superiority; p = 0.0280, MMRM; LS mean difference = -1.2, 90% CI 2-sided [-2.18 to -0.17], Standard Error of Mean 0.60
Statistical Analysis 49: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; [analysis description as in outcome 4, analysis 43]; Test type: Superiority; p = 0.0781, MMRM; LS mean difference = -0.9, 90% CI 2-sided [-1.98 to 0.15], Standard Error of Mean 0.64

11. Secondary Outcome: Change From Baseline in PP-NRS Score at Week 14 and 16
Description: as for outcome 8
Time Frame: Baseline, Week 14 and 16
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 26 | 24 | 23 | 20 | 27 | 27 | 21 | 23 | 18
Unit on a scale
  Change at Week 14: number analyzed (Participants) | 26 | 23 | 23 | 20 | 27 | 24 | 21 | 23 | 18
  Change at Week 14 | -0.4 (3.18) | -1.4 (1.64) | -1.8 (3.16) | -1.2 (2.52) | -1.1 (2.38) | -1.0 (2.93) | -1.1 (2.57) | -1.3 (2.31) | -0.1 (4.18)
  Change at Week 16: number analyzed (Participants) | 25 | 24 | 22 | 19 | 25 | 27 | 20 | 20 | 16
  Change at Week 16 | -0.6 (2.97) | -0.9 (1.82) | -1.2 (3.21) | -0.7 (2.02) | -1.0 (2.52) | -0.9 (2.99) | -1.0 (2.29) | -0.9 (2.25) | 0.4 (3.54)

12. Secondary Outcome: Absolute Psoriasis Symptom Inventory (PSI) Score at Baseline, Week 1, 2, 4, 6, 8, 10, 12, 14 and 16, Early Termination (ET), ET Follow-up Visit 1 and 2
Description: PSI was a self-administered 8-item questionnaire that measured the severity of psoriasis symptoms over the past 24 hours and the past 7 days. PSI included following 8 items: itch, pain, burning, stinging, cracking, scaling, flaking, and redness. Each item was rated on a scale from 0 to 4, where 0= not at all severe, 1= mild, 2= moderate, 3= severe and 4= very severe. Scores from all items were summed to give PSI score range from 0 (no severity) to 32 (maximum severity), higher PSI score indicated greater severity.
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10, 12, 14 and 16, ET (Prior to Week 12), ET Follow-up Visit 1 (2 weeks post ET) and 2 (4 weeks post ET)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 35 | 36 | 34 | 36 | 37 | 48 | 35 | 35 | 31
Unit on a scale
  Baseline: number analyzed (Participants) | 33 | 34 | 33 | 29 | 36 | 43 | 33 | 33 | 30
  Baseline | 14.2 (5.96) | 12.3 (7.18) | 13.2 (6.55) | 10.3 (5.00) | 12.3 (6.48) | 14.0 (6.60) | 13.0 (6.09) | 10.1 (5.70) | 16.6 (7.01)
  Week 1: number analyzed (Participants) | 35 | 36 | 34 | 36 | 37 | 47 | 35 | 34 | 29
  Week 1 | 11.2 (4.17) | 9.1 (5.85) | 9.7 (5.29) | 7.8 (4.23) | 8.9 (6.10) | 9.6 (4.86) | 9.5 (4.86) | 7.0 (4.96) | 9.7 (4.24)
  Week 2: number analyzed (Participants) | 35 | 36 | 33 | 35 | 35 | 48 | 35 | 35 | 31
  Week 2 | 10.3 (4.57) | 8.4 (5.07) | 9.2 (5.03) | 7.1 (4.01) | 8.2 (5.17) | 8.4 (4.52) | 9.1 (5.47) | 6.0 (4.30) | 8.4 (3.62)
  Week 4: number analyzed (Participants) | 32 | 31 | 27 | 33 | 34 | 46 | 29 | 31 | 31
  Week 4 | 11.6 (5.81) | 9.2 (5.25) | 9.9 (5.29) | 7.3 (3.97) | 8.1 (4.89) | 9.6 (6.96) | 7.9 (5.57) | 6.6 (4.60) | 8.3 (3.99)
  Week 6: number analyzed (Participants) | 32 | 30 | 25 | 31 | 28 | 38 | 27 | 27 | 27
  Week 6 | 11.6 (6.61) | 9.7 (5.79) | 10.4 (6.20) | 6.2 (3.79) | 7.6 (4.69) | 8.8 (5.96) | 6.1 (3.23) | 6.9 (5.06) | 8.2 (4.23)
  Week 8: number analyzed (Participants) | 30 | 31 | 26 | 31 | 26 | 36 | 24 | 28 | 27
  Week 8 | 11.3 (5.82) | 8.7 (5.87) | 9.7 (6.62) | 6.1 (3.73) | 7.0 (4.61) | 8.4 (5.46) | 7.2 (4.75) | 7.5 (4.92) | 8.0 (4.68)
  Week 10: number analyzed (Participants) | 29 | 28 | 25 | 29 | 28 | 31 | 24 | 28 | 24
  Week 10 | 11.7 (7.09) | 8.0 (6.29) | 9.5 (5.89) | 6.5 (3.66) | 6.4 (4.87) | 7.8 (4.92) | 6.7 (3.13) | 6.7 (4.60) | 9.5 (4.97)
  Week 12: number analyzed (Participants) | 29 | 29 | 26 | 29 | 27 | 31 | 23 | 28 | 25
  Week 12 | 11.7 (7.40) | 7.8 (6.41) | 9.7 (6.45) | 5.9 (3.38) | 6.2 (4.69) | 8.0 (5.13) | 6.1 (3.67) | 6.8 (5.14) | 8.3 (4.79)
  Week 14: number analyzed (Participants) | 28 | 25 | 24 | 24 | 27 | 27 | 23 | 25 | 23
  Week 14 | 14.3 (8.09) | 8.1 (6.37) | 8.9 (6.09) | 6.8 (5.00) | 9.2 (6.12) | 10.4 (5.98) | 11.2 (7.54) | 8.5 (6.04) | 11.5 (5.26)
  Week 16: number analyzed (Participants) | 27 | 27 | 23 | 24 | 25 | 30 | 22 | 22 | 19
  Week 16 | 14.0 (7.60) | 8.6 (6.30) | 9.8 (5.47) | 7.4 (5.03) | 8.9 (6.77) | 10.4 (6.18) | 11.5 (7.20) | 10.2 (6.82) | 11.9 (7.33)
  ET: number analyzed (Participants) | 3 | 3 | 5 | 3 | 4 | 6 | 6 | 4 | 3
  ET | 7.7 (4.04) | 13.0 (1.00) | 12.8 (6.76) | 13.3 (7.02) | 15.8 (11.73) | 18.7 (10.23) | 18.0 (11.87) | 11.0 (8.21) | 19.3 (8.14)
  ET follow-up visit 1: number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 2 | 1 | 1
  ET follow-up visit 1 | 7.0 (4.24) | 9.0 (NA) — Standard deviation could not be estimated due to insufficient number of participants with event. | 6.0 (4.24) | 4.0 (NA) — Standard deviation could not be estimated due to insufficient number of participants with event. | 2.0 (NA) — Standard deviation could not be estimated due to insufficient number of participants with event. | 19.0 (15.56) | 8.5 (2.12) | 4.0 (NA) — Standard deviation could not be estimated due to insufficient number of participants with event. | 7.0 (NA) — Standard deviation could not be estimated due to insufficient number of participants with event.
  ET follow-up visit 2: number analyzed (Participants) | 2 | 1 | 2 | 1 | 2 | 4 | 2 | 4 | 2
  ET follow-up visit 2 | 8.0 (5.66) | 7.0 (NA) — Standard deviation could not be estimated due to insufficient number of participants with event. | 4.5 (2.12) | 4.0 (NA) — Standard deviation could not be estimated due to insufficient number of participants with event. | 22.5 (9.19) | 17.8 (11.41) | 4.0 (0.00) | 13.0 (13.74) | 15.5 (10.61)

13. Secondary Outcome: Change From Baseline in PSI Score at Week 1, 2, 4, 6, 8, 10, 12, 14 and 16, ET, ET Follow-up Visit 1 and 2
Description: as for outcome 12
Time Frame: as for outcome 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 33 | 34 | 32 | 29 | 36 | 43 | 33 | 33 | 28
Unit on a scale
  Change at Week 1 | -3.3 (4.94) | -2.8 (3.35) | -3.0 (3.84) | -2.6 (2.95) | -3.4 (4.17) | -3.9 (5.00) | -3.7 (3.49) | -3.4 (3.18) | -6.6 (4.80)
  Change at Week 2: number analyzed (Participants) | 33 | 33 | 31 | 29 | 34 | 43 | 33 | 33 | 28
  Change at Week 2 | -4.0 (5.46) | -3.9 (4.91) | -4.1 (4.36) | -3.1 (3.63) | -3.8 (4.62) | -5.1 (5.85) | -4.2 (3.91) | -4.3 (4.12) | -7.8 (5.37)
  Change at Week 4: number analyzed (Participants) | 30 | 28 | 26 | 27 | 33 | 40 | 27 | 29 | 25
  Change at Week 4 | -3.0 (6.33) | -3.4 (5.09) | -3.5 (5.12) | -2.6 (3.91) | -4.1 (4.55) | -3.9 (6.50) | -4.6 (5.44) | -3.7 (4.57) | -6.5 (5.44)
  Change at Week 6: number analyzed (Participants) | 30 | 28 | 24 | 25 | 28 | 32 | 25 | 26 | 22
  Change at Week 6 | -3.5 (7.09) | -3.1 (5.30) | -2.0 (6.20) | -3.5 (5.22) | -4.0 (4.64) | -5.1 (7.40) | -6.3 (5.05) | -3.4 (4.60) | -6.5 (5.75)
  Change at Week 8: number analyzed (Participants) | 28 | 28 | 25 | 25 | 26 | 30 | 22 | 27 | 22
  Change at Week 8 | -4.1 (7.20) | -3.5 (4.60) | -3.2 (6.56) | -3.7 (5.01) | -4.1 (5.01) | -5.2 (8.12) | -5.8 (5.35) | -3.2 (4.90) | -7.0 (6.64)
  Change at Week 10: number analyzed (Participants) | 27 | 25 | 24 | 23 | 28 | 26 | 23 | 27 | 20
  Change at Week 10 | -4.0 (7.57) | -4.0 (4.90) | -3.4 (6.24) | -3.3 (6.12) | -5.3 (5.69) | -5.5 (8.08) | -5.1 (5.12) | -3.9 (4.82) | -5.8 (7.62)
  Change at Week 12: number analyzed (Participants) | 27 | 26 | 25 | 23 | 27 | 28 | 22 | 27 | 19
  Change at Week 12 | -3.8 (7.74) | -4.1 (4.98) | -3.2 (5.63) | -3.7 (6.13) | -5.2 (6.04) | -5.0 (8.15) | -5.2 (4.82) | -3.7 (5.67) | -6.6 (7.82)
  Change at Week 14: number analyzed (Participants) | 26 | 23 | 23 | 20 | 27 | 24 | 21 | 24 | 18
  Change at Week 14 | -0.7 (7.86) | -2.9 (4.68) | -4.4 (7.49) | -3.1 (6.87) | -2.2 (5.49) | -3.5 (7.87) | -1.4 (5.53) | -2.3 (4.98) | -2.9 (7.98)
  Change at Week 16: number analyzed (Participants) | 25 | 24 | 22 | 19 | 25 | 27 | 20 | 21 | 16
  Change at Week 16 | -0.9 (7.61) | -2.4 (5.02) | -3.2 (6.37) | -2.4 (7.27) | -2.1 (6.05) | -2.6 (7.12) | -0.8 (4.29) | -0.8 (5.28) | -2.7 (8.40)
  Change at ET: number analyzed (Participants) | 3 | 3 | 4 | 3 | 4 | 6 | 5 | 3 | 2
  Change at ET | -2.7 (2.52) | 0.7 (6.11) | -1.0 (8.29) | 0.3 (2.08) | -1.3 (6.85) | 0.7 (5.16) | 1.8 (7.40) | -4.0 (3.00) | -5.0 (1.41)
  Change at ET Follow-up Visit 1: number analyzed (Participants) | 2 | 1 | 2 | 1 | 1 | 2 | 2 | 1 | 1
  Change at ET Follow-up Visit 1 | -2.5 (0.71) | -9.0 (NA) — Standard deviation could not be estimated due to insufficient number of participants with event. | -5.0 (7.07) | -4.0 (NA) — Standard deviation could not be estimated due to insufficient number of participants with event. | -3.0 (NA) — Standard deviation could not be estimated due to insufficient number of participants with event. | 2.0 (9.90) | -2.5 (0.71) | -7.0 (NA) — Standard deviation could not be estimated due to insufficient number of participants with event. | -9.0 (NA) — Standard deviation could not be estimated due to insufficient number of participants with event.
  Change at ET Follow-up Visit 2: number analyzed (Participants) | 2 | 1 | 2 | 1 | 2 | 4 | 2 | 4 | 2
  Change at ET Follow-up Visit 2 | -1.5 (2.12) | -11.0 (NA) — Standard deviation could not be estimated due to insufficient number of participants with event. | -6.5 (4.95) | -4.0 (NA) — Standard deviation could not be estimated due to insufficient number of participants with event. | 6.5 (9.19) | 0.8 (7.14) | -11.0 (4.24) | -0.3 (8.26) | -1.0 (9.90)

14. Secondary Outcome: Percentage of Participants With PGA Score Clear (0) or Almost Clear (1) and >=2 Points Improvement From Baseline at Week 1, 2, 4, 6, 8, 10, 14, and 16
Description: as for outcome 2
Time Frame: Baseline, Week 1, 2, 4, 6, 8, 10, 14, and 16
Population: as for outcome 5
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 36 | 37 | 37 | 36 | 37 | 49 | 36 | 35 | 38
Percentage of participants
  Week 1 | 2.8 [0.3 to 11.6] | 2.7 [0.3 to 11.2] | 2.7 [0.3 to 11.2] | 0 [0.0 to 7.5] | 0 [0.0 to 7.3] | 0 [0.0 to 5.5] | 0 [0.0 to 7.5] | 5.7 [1.5 to 16.4] | 5.3 [1.4 to 15.0]
  Week 2 | 2.8 [0.3 to 11.6] | 0 [0.0 to 7.3] | 0 [0.0 to 7.3] | 2.8 [0.3 to 11.6] | 2.7 [0.3 to 11.2] | 2.0 [0.2 to 8.4] | 0 [0.0 to 7.5] | 5.7 [1.5 to 16.4] | 10.5 [4.7 to 21.6]
  Week 4 | 5.6 [1.5 to 15.9] | 5.4 [1.4 to 15.5] | 0 [0.0 to 7.3] | 5.6 [1.5 to 15.9] | 5.4 [1.4 to 15.5] | 8.2 [3.6 to 16.5] | 8.3 [3.1 to 18.9] | 11.4 [5.1 to 23.6] | 21.1 [10.9 to 33.3]
  Week 6 | 8.3 [3.1 to 18.9] | 5.4 [1.4 to 15.5] | 2.7 [0.3 to 11.2] | 8.3 [3.1 to 18.9] | 13.5 [6.7 to 24.8] | 8.2 [3.6 to 16.5] | 8.3 [3.1 to 18.9] | 5.7 [1.5 to 16.4] | 13.2 [6.5 to 24.3]
  Week 8 | 11.1 [4.9 to 22.9] | 5.4 [1.4 to 15.5] | 5.4 [1.4 to 15.5] | 2.8 [0.3 to 11.6] | 10.8 [4.8 to 22.2] | 6.1 [2.3 to 14.8] | 13.9 [6.9 to 25.4] | 5.7 [1.5 to 16.4] | 18.4 [10.1 to 30.9]
  Week 10 | 8.3 [3.1 to 18.9] | 5.4 [1.4 to 15.5] | 8.1 [3.0 to 18.5] | 8.3 [3.1 to 18.9] | 16.2 [7.3 to 29.3] | 16.3 [8.4 to 27.1] | 16.7 [7.5 to 30.2] | 8.6 [3.2 to 19.3] | 13.2 [6.5 to 24.3]
  Week 14: number analyzed (Participants) | 36 | 37 | 36 | 35 | 37 | 48 | 34 | 34 | 37
  Week 14 | 2.8 [0.3 to 11.6] | 13.5 [6.7 to 24.8] | 5.6 [1.5 to 15.9] | 8.6 [3.2 to 19.3] | 13.5 [6.7 to 24.8] | 6.3 [2.3 to 15.1] | 8.8 [3.3 to 19.7] | 11.8 [5.2 to 24.3] | 8.1 [3.0 to 18.5]
  Week 16: number analyzed (Participants) | 36 | 35 | 35 | 35 | 37 | 49 | 34 | 34 | 37
  Week 16 | 5.6 [1.5 to 15.9] | 11.4 [5.1 to 23.6] | 8.6 [3.2 to 19.3] | 14.3 [7.1 to 26.0] | 16.2 [7.3 to 29.3] | 8.2 [3.6 to 16.5] | 14.7 [7.3 to 26.9] | 11.8 [5.2 to 24.3] | 16.2 [7.3 to 29.3]
Statistical Analysis 1: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 1; Test type: Superiority; p = 0.4216, Chan and Zhang method; Risk Difference (RD) = -0.1, 90% CI 2-sided [-9.4 to 9.1]
Statistical Analysis 2: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 1; Test type: Superiority; p = 0.4216, Chan and Zhang method; Risk Difference (RD) = -0.1, 90% CI 2-sided [-9.4 to 9.1]
Statistical Analysis 3: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 1; Test type: Superiority; p = 0.7362, Chan and Zhang method; Risk Difference (RD) = -2.8, 90% CI 2-sided [-12.5 to 5.0]
Statistical Analysis 4: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 1; Test type: Superiority; p = 0.7417, Chan and Zhang method; Risk Difference (RD) = -2.8, 90% CI 2-sided [-12.5 to 4.7]
Statistical Analysis 5: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 1; Test type: Superiority; p = 0.5000, Chan and Zhang method; Risk Difference (RD) = 0.0, 90% CI 2-sided [-5.9 to 8.0]
Statistical Analysis 6: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 1; Test type: Superiority; p = 0.0714, Chan and Zhang method; Risk Difference (RD) = 5.7, 90% CI 2-sided [-0.8 to 16.9]
Statistical Analysis 7: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 1; Test type: Superiority; p = 0.0813, Chan and Zhang method; Risk Difference (RD) = 5.3, 90% CI 2-sided [-1.1 to 15.7]
Statistical Analysis 8: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 2; Test type: Superiority; p = 0.7417, Chan and Zhang method; Risk Difference (RD) = -2.8, 90% CI 2-sided [-12.5 to 4.7]
Statistical Analysis 9: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 2; Test type: Superiority; p = 0.7417, Chan and Zhang method; Risk Difference (RD) = -2.8, 90% CI 2-sided [-12.5 to 4.7]
Statistical Analysis 10: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 2; Test type: Superiority; p = 0.5000, Chan and Zhang method; Risk Difference (RD) = 0.0, 90% CI 2-sided [-9.6 to 9.6]
Statistical Analysis 11: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 2; Test type: Superiority; p = 0.4216, Chan and Zhang method; Risk Difference (RD) = -0.1, 90% CI 2-sided [-9.4 to 9.1]
Statistical Analysis 12: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 2; Test type: Superiority; p = 0.6894, Chan and Zhang method; Risk Difference (RD) = -2.0, 90% CI 2-sided [-9.4 to 5.9]
Statistical Analysis 13: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 2; Test type: Superiority; p = 0.2518, Chan and Zhang method; Risk Difference (RD) = 3.7, 90% CI 2-sided [-4.2 to 14.3]
Statistical Analysis 14: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 2; Test type: Superiority; p = 0.0565, Chan and Zhang method; Risk Difference (RD) = 8.5, 90% CI 2-sided [-0.3 to 20.3]
Statistical Analysis 15: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 4; Test type: Superiority; p = 0.4446, Chan and Zhang method; Risk Difference (RD) = -0.2, 90% CI 2-sided [-11.0 to 11.0]
Statistical Analysis 16: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 4; Test type: Superiority; p = 0.9001, Chan and Zhang method; Risk Difference (RD) = -5.6, 90% CI 2-sided [-16.5 to 1.9]
Statistical Analysis 17: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 4; Test type: Superiority; p = 0.5000, Chan and Zhang method; Risk Difference (RD) = 0.0, 90% CI 2-sided [-11.0 to 11.0]
Statistical Analysis 18: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 4; Test type: Superiority; p = 0.4446, Chan and Zhang method; Risk Difference (RD) = -0.2, 90% CI 2-sided [-11.0 to 11.0]
Statistical Analysis 19: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 4; Test type: Superiority; p = 0.5054, Chan and Zhang method; Risk Difference (RD) = 0.2, 90% CI 2-sided [-10.5 to 12.5]
Statistical Analysis 20: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 4; Test type: Superiority; p = 0.3401, Chan and Zhang method; Risk Difference (RD) = 3.3, 90% CI 2-sided [-8.2 to 16.9]
Statistical Analysis 21: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 4; Test type: Superiority; p = 0.0489, Chan and Zhang method; Risk Difference (RD) = 12.9, 90% CI 2-sided [0.1 to 27.5]
Statistical Analysis 22: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 6; Test type: Superiority; p = 0.6349, Chan and Zhang method; Risk Difference (RD) = -2.9, 90% CI 2-sided [-14.8 to 8.4]
Statistical Analysis 23: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 6; Test type: Superiority; p = 0.8253, Chan and Zhang method; Risk Difference (RD) = -5.6, 90% CI 2-sided [-17.2 to 4.4]
Statistical Analysis 24: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 6; Test type: Superiority; p = 0.5000, Chan and Zhang method; Risk Difference (RD) = 0.0, 90% CI 2-sided [-12.5 to 12.5]
Statistical Analysis 25: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 6; Test type: Superiority; p = 0.2709, Chan and Zhang method; Risk Difference (RD) = 5.2, 90% CI 2-sided [-8.3 to 19.1]
Statistical Analysis 26: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 6; Test type: Superiority; p = 0.5054, Chan and Zhang method; Risk Difference (RD) = 0.2, 90% CI 2-sided [-10.5 to 12.5]
Statistical Analysis 27: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 6; Test type: Superiority; p = 0.6319, Chan and Zhang method; Risk Difference (RD) = -2.4, 90% CI 2-sided [-12.9 to 9.3]
Statistical Analysis 28: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 6; Test type: Superiority; p = 0.3199, Chan and Zhang method; Risk Difference (RD) = 5.0, 90% CI 2-sided [-6.4 to 18.1]
Statistical Analysis 29: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 8; Test type: Superiority; p = 0.7306, Chan and Zhang method; Risk Difference (RD) = -5.7, 90% CI 2-sided [-19.1 to 6.1]
Statistical Analysis 30: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 8; Test type: Superiority; p = 0.7306, Chan and Zhang method; Risk Difference (RD) = -5.7, 90% CI 2-sided [-19.1 to 6.1]
Statistical Analysis 31: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 8; Test type: Superiority; p = 0.8808, Chan and Zhang method; Risk Difference (RD) = -8.3, 90% CI 2-sided [-20.6 to 2.7]
Statistical Analysis 32: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 8; Test type: Superiority; p = 0.4644, Chan and Zhang method; Risk Difference (RD) = -0.3, 90% CI 2-sided [-13.7 to 13.7]
Statistical Analysis 33: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 8; Test type: Superiority; p = 0.1534, Chan and Zhang method; Risk Difference (RD) = 7.8, 90% CI 2-sided [-3.4 to 20.9]
Statistical Analysis 34: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 8; Test type: Superiority; p = 0.4867, Chan and Zhang method; Risk Difference (RD) = -0.4, 90% CI 2-sided [-10.0 to 11.4]
Statistical Analysis 35: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 8; Test type: Superiority; p = 0.0435, Chan and Zhang method; Risk Difference (RD) = 12.3, 90% CI 2-sided [0.4 to 25.9]
Statistical Analysis 36: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 10; Test type: Superiority; p = 0.6349, Chan and Zhang method; Risk Difference (RD) = -2.9, 90% CI 2-sided [-14.8 to 8.4]
Statistical Analysis 37: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 10; Test type: Superiority; p = 0.4565, Chan and Zhang method; Risk Difference (RD) = -0.2, 90% CI 2-sided [-12.6 to 12.5]
Statistical Analysis 38: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 10; Test type: Superiority; p = 0.5000, Chan and Zhang method; Risk Difference (RD) = 0.0, 90% CI 2-sided [-12.5 to 12.5]
Statistical Analysis 39: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 10; Test type: Superiority; p = 0.1765, Chan and Zhang method; Risk Difference (RD) = 7.9, 90% CI 2-sided [-5.7 to 21.8]
Statistical Analysis 40: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 10; Test type: Superiority; p = 0.5013, Chan and Zhang method; Risk Difference (RD) = 0.3, 90% CI 2-sided [-14.0 to 15.2]
Statistical Analysis 41: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 10; Test type: Superiority; p = 0.7969, Chan and Zhang method; Risk Difference (RD) = -7.8, 90% CI 2-sided [-20.7 to 5.9]
Statistical Analysis 42: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 10; Test type: Superiority; p = 0.6424, Chan and Zhang method; Risk Difference (RD) = -3.2, 90% CI 2-sided [-16.4 to 10.6]
Statistical Analysis 43: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 14; Test type: Superiority; p = 0.0620, Chan and Zhang method; Risk Difference (RD) = 10.7, 90% CI 2-sided [-0.7 to 23.6]
Statistical Analysis 44: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 14; Test type: Superiority; p = 0.3402, Chan and Zhang method; Risk Difference (RD) = 2.8, 90% CI 2-sided [-7.0 to 13.4]
Statistical Analysis 45: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 14; Test type: Superiority; p = 0.1743, Chan and Zhang method; Risk Difference (RD) = 5.8, 90% CI 2-sided [-4.5 to 17.6]
Statistical Analysis 46: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 14; Test type: Superiority; p = 0.0620, Chan and Zhang method; Risk Difference (RD) = 10.7, 90% CI 2-sided [-0.7 to 23.6]
Statistical Analysis 47: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 14; Test type: Superiority; p = 0.3534, Chan and Zhang method; Risk Difference (RD) = 2.6, 90% CI 2-sided [-7.8 to 15.4]
Statistical Analysis 48: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 14; Test type: Superiority; p = 0.2508, Chan and Zhang method; Risk Difference (RD) = 5.5, 90% CI 2-sided [-5.5 to 18.8]
Statistical Analysis 49: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 14; Test type: Superiority; p = 0.4238, Chan and Zhang method; Risk Difference (RD) = 1.9, 90% CI 2-sided [-8.2 to 13.6]
Statistical Analysis 50: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 16; Test type: Superiority; p = 0.2696, Chan and Zhang method; Risk Difference (RD) = 5.9, 90% CI 2-sided [-6.2 to 19.3]
Statistical Analysis 51: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 16; Test type: Superiority; p = 0.3648, Chan and Zhang method; Risk Difference (RD) = 3.0, 90% CI 2-sided [-8.6 to 15.3]
Statistical Analysis 52: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 16; Test type: Superiority; p = 0.1267, Chan and Zhang method; Risk Difference (RD) = 8.7, 90% CI 2-sided [-3.8 to 22.2]
Statistical Analysis 53: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 16; Test type: Superiority; p = 0.0832, Chan and Zhang method; Risk Difference (RD) = 10.7, 90% CI 2-sided [-2.5 to 24.4]
Statistical Analysis 54: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 16; Test type: Superiority; p = 0.2099, Chan and Zhang method; Risk Difference (RD) = 6.5, 90% CI 2-sided [-5.7 to 21.3]
Statistical Analysis 55: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 16; Test type: Superiority; p = 0.3474, Chan and Zhang method; Risk Difference (RD) = 3.6, 90% CI 2-sided [-8.0 to 17.4]
Statistical Analysis 56: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 16; Test type: Superiority; p = 0.2124, Chan and Zhang method; Risk Difference (RD) = 8.1, 90% CI 2-sided [-4.0 to 21.6]

15. Secondary Outcome: Percentage of Participants Who Achieved PSI Score of 0 (Not at All) or 1 (Mild) on All Items at Week 1, 2, 4, 6, 8, 10, 12, 14, and 16
Description: as for outcome 12
Time Frame: Week 1, 2, 4, 6, 8, 10, 12, 14, and 16
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 35 | 36 | 34 | 36 | 37 | 48 | 35 | 35 | 31
Percentage of participants
  Week 1: number analyzed (Participants) | 35 | 36 | 34 | 36 | 37 | 47 | 35 | 34 | 29
  Week 1 | 5.7 [1.5 to 16.4] | 19.4 [10.7 to 32.8] | 11.8 [5.2 to 24.3] | 22.2 [11.6 to 35.3] | 13.5 [6.7 to 24.8] | 19.1 [11.2 to 30.3] | 11.4 [5.1 to 23.6] | 26.5 [15.9 to 40.5] | 24.1 [13.4 to 38.5]
  Week 2: number analyzed (Participants) | 35 | 36 | 33 | 35 | 35 | 48 | 35 | 35 | 31
  Week 2 | 8.6 [3.2 to 19.3] | 22.2 [11.6 to 35.3] | 18.2 [8.2 to 31.3] | 34.3 [22.0 to 47.8] | 31.4 [19.3 to 44.8] | 20.8 [11.8 to 31.5] | 25.7 [15.4 to 39.2] | 31.4 [19.3 to 44.8] | 32.3 [18.7 to 48.2]
  Week 4: number analyzed (Participants) | 32 | 31 | 27 | 33 | 34 | 46 | 29 | 31 | 31
  Week 4 | 15.6 [7.8 to 28.7] | 29.0 [17.6 to 45.0] | 29.6 [15.7 to 45.3] | 48.5 [34.4 to 63.9] | 38.2 [24.3 to 53.8] | 26.1 [15.8 to 37.7] | 31.0 [18.9 to 46.3] | 51.6 [36.8 to 67.3] | 35.5 [21.3 to 51.8]
  Week 6: number analyzed (Participants) | 32 | 30 | 25 | 31 | 28 | 38 | 27 | 27 | 27
  Week 6 | 18.8 [8.5 to 32.0] | 26.7 [14.0 to 41.6] | 32.0 [17.0 to 50.0] | 54.8 [39.9 to 70.3] | 42.9 [28.4 to 60.0] | 31.6 [19.9 to 45.9] | 66.7 [50.0 to 79.6] | 48.1 [32.6 to 65.3] | 33.3 [20.4 to 50.0]
  Week 8: number analyzed (Participants) | 30 | 31 | 26 | 31 | 26 | 36 | 24 | 28 | 27
  Week 8 | 23.3 [12.9 to 37.6] | 35.5 [21.3 to 51.8] | 46.2 [29.9 to 63.8] | 67.7 [51.8 to 81.3] | 50.0 [34.2 to 65.8] | 41.7 [29.0 to 56.0] | 62.5 [44.7 to 77.9] | 35.7 [20.8 to 52.7] | 59.3 [41.7 to 75.2]
  Week 10: number analyzed (Participants) | 29 | 28 | 25 | 29 | 28 | 31 | 24 | 28 | 24
  Week 10 | 31.0 [18.9 to 46.3] | 42.9 [28.4 to 60.0] | 40.0 [24.6 to 58.3] | 62.1 [46.3 to 77.1] | 64.3 [47.3 to 79.2] | 45.2 [29.7 to 60.1] | 50.0 [31.9 to 68.1] | 46.4 [31.0 to 63.4] | 33.3 [17.8 to 52.1]
  Week 12: number analyzed (Participants) | 29 | 29 | 26 | 29 | 27 | 31 | 23 | 28 | 25
  Week 12 | 24.1 [13.4 to 38.5] | 51.7 [35.2 to 68.0] | 50.0 [34.2 to 65.8] | 62.1 [46.3 to 77.1] | 55.6 [38.2 to 70.9] | 35.5 [21.3 to 51.8] | 56.5 [38.1 to 72.7] | 46.4 [31.0 to 63.4] | 36.0 [21.4 to 54.4]
  Week 14: number analyzed (Participants) | 28 | 25 | 24 | 24 | 27 | 27 | 23 | 25 | 23
  Week 14 | 7.1 [1.9 to 20.1] | 44.0 [27.0 to 61.1] | 45.8 [28.2 to 63.0] | 54.2 [37.0 to 71.8] | 37.0 [22.1 to 54.7] | 25.9 [14.5 to 41.7] | 30.4 [17.3 to 47.9] | 36.0 [21.4 to 54.4] | 17.4 [7.8 to 33.5]
  Week 16: number analyzed (Participants) | 27 | 27 | 23 | 24 | 25 | 30 | 22 | 22 | 19
  Week 16 | 7.4 [2.0 to 20.4] | 44.4 [29.1 to 61.8] | 30.4 [17.3 to 47.9] | 54.2 [37.0 to 71.8] | 52.0 [36.0 to 69.3] | 36.7 [22.1 to 52.4] | 18.2 [8.2 to 35.3] | 22.7 [11.5 to 39.5] | 31.6 [15.1 to 53.0]
Statistical Analysis 1: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 1; Test type: Superiority; p = 0.0544, Chan and Zhang method; Risk Difference (RD) = 13.7, 90% CI 2-sided [-0.3 to 27.9]
Statistical Analysis 2: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 1; Test type: Superiority; p = 0.2697, Chan and Zhang method; Risk Difference (RD) = 6.1, 90% CI 2-sided [-6.3 to 19.6]
Statistical Analysis 3: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 1; Test type: Superiority; p = 0.0286, Chan and Zhang method; Risk Difference (RD) = 16.5, 90% CI 2-sided [2.0 to 31.0]
Statistical Analysis 4: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 1; Test type: Superiority; p = 0.1512, Chan and Zhang method; Risk Difference (RD) = 7.8, 90% CI 2-sided [-4.7 to 20.8]
Statistical Analysis 5: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 1; Test type: Superiority; p = 0.7900, Chan and Zhang method; Risk Difference (RD) = -7.7, 90% CI 2-sided [-21.9 to 7.4]
Statistical Analysis 6: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 1; Test type: Superiority; p = 0.3137, Chan and Zhang method; Risk Difference (RD) = 7.3, 90% CI 2-sided [-8.5 to 24.0]
Statistical Analysis 7: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 1; Test type: Superiority; p = 0.3789, Chan and Zhang method; Risk Difference (RD) = 5.0, 90% CI 2-sided [-10.9 to 22.6]
Statistical Analysis 8: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 2; Test type: Superiority; p = 0.0636, Chan and Zhang method; Risk Difference (RD) = 13.7, 90% CI 2-sided [-1.0 to 28.5]
Statistical Analysis 9: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 2; Test type: Superiority; p = 0.1435, Chan and Zhang method; Risk Difference (RD) = 9.6, 90% CI 2-sided [-4.9 to 24.5]
Statistical Analysis 10: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 2; Test type: Superiority; p = 0.0058, Chan and Zhang method; Risk Difference (RD) = 25.7, 90% CI 2-sided [8.9 to 42.4]
Statistical Analysis 11: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 2; Test type: Superiority; p = 0.0112, Chan and Zhang method; Risk Difference (RD) = 22.9, 90% CI 2-sided [6.5 to 38.9]
Statistical Analysis 12: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 2; Test type: Superiority; p = 0.3349, Chan and Zhang method; Risk Difference (RD) = 4.9, 90% CI 2-sided [-10.8 to 21.3]
Statistical Analysis 13: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 2; Test type: Superiority; p = 0.2065, Chan and Zhang method; Risk Difference (RD) = 10.6, 90% CI 2-sided [-6.1 to 27.7]
Statistical Analysis 14: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 2; Test type: Superiority; p = 0.1871, Chan and Zhang method; Risk Difference (RD) = 11.4, 90% CI 2-sided [-5.6 to 29.1]
Statistical Analysis 15: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 4; Test type: Superiority; p = 0.1245, Chan and Zhang method; Risk Difference (RD) = 13.4, 90% CI 2-sided [-4.9 to 31.4]
Statistical Analysis 16: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 4; Test type: Superiority; p = 0.1280, Chan and Zhang method; Risk Difference (RD) = 14.0, 90% CI 2-sided [-4.7 to 33.7]
Statistical Analysis 17: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 4; Test type: Superiority; p = 0.0030, Chan and Zhang method; Risk Difference (RD) = 32.9, 90% CI 2-sided [12.4 to 50.5]
Statistical Analysis 18: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 4; Test type: Superiority; p = 0.0235, Chan and Zhang method; Risk Difference (RD) = 22.6, 90% CI 2-sided [3.1 to 40.6]
Statistical Analysis 19: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 4; Test type: Superiority; p = 0.3728, Chan and Zhang method; Risk Difference (RD) = 4.9, 90% CI 2-sided [-13.6 to 24.1]
Statistical Analysis 20: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 4; Test type: Superiority; p = 0.0153, Chan and Zhang method; Risk Difference (RD) = 25.5, 90% CI 2-sided [4.0 to 43.6]
Statistical Analysis 21: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 4; Test type: Superiority; p = 0.2543, Chan and Zhang method; Risk Difference (RD) = 9.4, 90% CI 2-sided [-8.8 to 27.8]
Statistical Analysis 22: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 6; Test type: Superiority; p = 0.2785, Chan and Zhang method; Risk Difference (RD) = 7.9, 90% CI 2-sided [-10.2 to 26.4]
Statistical Analysis 23: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 6; Test type: Superiority; p = 0.1434, Chan and Zhang method; Risk Difference (RD) = 13.3, 90% CI 2-sided [-7.4 to 33.7]
Statistical Analysis 24: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 6; Test type: Superiority; p = 0.0015, Chan and Zhang method; Risk Difference (RD) = 36.1, 90% CI 2-sided [12.8 to 54.1]
Statistical Analysis 25: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 6; Test type: Superiority; p = 0.0242, Chan and Zhang method; Risk Difference (RD) = 24.1, 90% CI 2-sided [3.4 to 43.9]
Statistical Analysis 26: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 6; Test type: Superiority; p = 0.0037, Chan and Zhang method; Risk Difference (RD) = 35.1, 90% CI 2-sided [10.0 to 54.1]
Statistical Analysis 27: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 6; Test type: Superiority; p = 0.1037, Chan and Zhang method; Risk Difference (RD) = 16.6, 90% CI 2-sided [-4.9 to 36.7]
Statistical Analysis 28: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 6; Test type: Superiority; p = 0.4607, Chan and Zhang method; Risk Difference (RD) = 1.8, 90% CI 2-sided [-17.7 to 22.5]
Statistical Analysis 29: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 8; Test type: Superiority; p = 0.1725, Chan and Zhang method; Risk Difference (RD) = 12.2, 90% CI 2-sided [-8.0 to 31.9]
Statistical Analysis 30: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 8; Test type: Superiority; p = 0.0451, Chan and Zhang method; Risk Difference (RD) = 22.8, 90% CI 2-sided [0.2 to 43.6]
Statistical Analysis 31: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 8; Test type: Superiority; p = 0.0003, Chan and Zhang method; Risk Difference (RD) = 44.4, 90% CI 2-sided [21.3 to 62.9]
Statistical Analysis 32: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 8; Test type: Superiority; p = 0.0239, Chan and Zhang method; Risk Difference (RD) = 26.7, 90% CI 2-sided [3.8 to 47.6]
Statistical Analysis 33: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 8; Test type: Superiority; p = 0.0643, Chan and Zhang method; Risk Difference (RD) = 20.8, 90% CI 2-sided [-2.1 to 41.2]
Statistical Analysis 34: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 8; Test type: Superiority; p = 0.6676, Chan and Zhang method; Risk Difference (RD) = -6.0, 90% CI 2-sided [-25.9 to 15.9]
Statistical Analysis 35: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 8; Test type: Superiority; p = 0.0898, Chan and Zhang method; Risk Difference (RD) = 17.6, 90% CI 2-sided [-4.2 to 37.8]
Statistical Analysis 36: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 10; Test type: Superiority; p = 0.2707, Chan and Zhang method; Risk Difference (RD) = 11.8, 90% CI 2-sided [-10.1 to 32.9]
Statistical Analysis 37: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 10; Test type: Superiority; p = 0.2981, Chan and Zhang method; Risk Difference (RD) = 9.0, 90% CI 2-sided [-14.2 to 31.0]
Statistical Analysis 38: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 10; Test type: Superiority; p = 0.0110, Chan and Zhang method; Risk Difference (RD) = 31.0, 90% CI 2-sided [8.0 to 51.4]
Statistical Analysis 39: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 10; Test type: Superiority; p = 0.0083, Chan and Zhang method; Risk Difference (RD) = 33.3, 90% CI 2-sided [9.1 to 53.2]
Statistical Analysis 40: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 10; Test type: Superiority; p = 0.4217, Chan and Zhang method; Risk Difference (RD) = 4.8, 90% CI 2-sided [-18.3 to 27.5]
Statistical Analysis 41: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 10; Test type: Superiority; p = 0.5152, Chan and Zhang method; Risk Difference (RD) = 1.3, 90% CI 2-sided [-20.8 to 23.2]
Statistical Analysis 42: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 10; Test type: Superiority; p = 0.7002, Chan and Zhang method; Risk Difference (RD) = -11.8, 90% CI 2-sided [-33.1 to 11.7]
Statistical Analysis 43: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 12; Test type: Superiority; p = 0.0169, Chan and Zhang method; Risk Difference (RD) = 27.6, 90% CI 2-sided [5.2 to 47.9]
Statistical Analysis 44: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 12; Test type: Superiority; p = 0.0283, Chan and Zhang method; Risk Difference (RD) = 25.9, 90% CI 2-sided [3.2 to 46.2]
Statistical Analysis 45: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 12; Test type: Superiority; p = 0.0020, Chan and Zhang method; Risk Difference (RD) = 37.9, 90% CI 2-sided [14.3 to 57.1]
Statistical Analysis 46: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 12; Test type: Superiority; p = 0.0095, Chan and Zhang method; Risk Difference (RD) = 31.4, 90% CI 2-sided [8.4 to 51.5]
Statistical Analysis 47: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 12; Test type: Superiority; p = 0.0798, Chan and Zhang method; Risk Difference (RD) = 21.0, 90% CI 2-sided [-2.7 to 42.6]
Statistical Analysis 48: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 12; Test type: Superiority; p = 0.2848, Chan and Zhang method; Risk Difference (RD) = 10.9, 90% CI 2-sided [-11.3 to 31.8]
Statistical Analysis 49: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 12; Test type: Superiority; p = 0.5062, Chan and Zhang method; Risk Difference (RD) = 0.5, 90% CI 2-sided [-21.1 to 23.1]
Statistical Analysis 50: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 14; Test type: Superiority; p = 0.0012, Chan and Zhang method; Risk Difference (RD) = 36.9, 90% CI 2-sided [16.7 to 55.3]
Statistical Analysis 51: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 14; Test type: Superiority; p = 0.0007, Chan and Zhang method; Risk Difference (RD) = 38.7, 90% CI 2-sided [17.3 to 57.4]
Statistical Analysis 52: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 14; Test type: Superiority; p = 0.0001, Chan and Zhang method; Risk Difference (RD) = 47.0, 90% CI 2-sided [24.6 to 65.1]
Statistical Analysis 53: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 14; Test type: Superiority; p = 0.0039, Chan and Zhang method; Risk Difference (RD) = 29.9, 90% CI 2-sided [9.5 to 48.7]
Statistical Analysis 54: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 14; Test type: Superiority; p = 0.3895, Chan and Zhang method; Risk Difference (RD) = 4.5, 90% CI 2-sided [-17.5 to 26.5]
Statistical Analysis 55: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 14; Test type: Superiority; p = 0.2793, Chan and Zhang method; Risk Difference (RD) = 10.1, 90% CI 2-sided [-11.8 to 31.8]
Statistical Analysis 56: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 14; Test type: Superiority; p = 0.7027, Chan and Zhang method; Risk Difference (RD) = -8.5, 90% CI 2-sided [-28.4 to 12.2]
Statistical Analysis 57: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.1% QD; Week 16; Test type: Superiority; p = 0.0009, Chan and Zhang method; Risk Difference (RD) = 37.0, 90% CI 2-sided [15.4 to 55.2]
Statistical Analysis 58: Comparison: Vehicle Once Daily (QD) vs PF-06700841 0.3% QD; Week 16; Test type: Superiority; p = 0.0205, Chan and Zhang method; Risk Difference (RD) = 23.0, 90% CI 2-sided [4.1 to 43.2]
Statistical Analysis 59: Comparison: Vehicle Once Daily (QD) vs PF-06700841 1.0% QD; Week 16; Test type: Superiority; p = 0.0001, Chan and Zhang method; Risk Difference (RD) = 46.8, 90% CI 2-sided [24.6 to 65.7]
Statistical Analysis 60: Comparison: Vehicle Once Daily (QD) vs PF-06700841 3.0% QD; Week 16; Test type: Superiority; p = 0.0002, Chan and Zhang method; Risk Difference (RD) = 44.6, 90% CI 2-sided [21.5 to 62.9]
Statistical Analysis 61: Comparison: Pooled Vehicle BID vs PF-06700841 0.3% BID; Week 16; Test type: Superiority; p = 0.9209, Chan and Zhang method; Risk Difference (RD) = -18.5, 90% CI 2-sided [-38.3 to 3.2]
Statistical Analysis 62: Comparison: Pooled Vehicle BID vs PF-06700841 1.0% BID; Week 16; Test type: Superiority; p = 0.7930, Chan and Zhang method; Risk Difference (RD) = -13.9, 90% CI 2-sided [-34.4 to 8.7]
Statistical Analysis 63: Comparison: Pooled Vehicle BID vs PF-06700841 3.0% BID; Week 16; Test type: Superiority; p = 0.6156, Chan and Zhang method; Risk Difference (RD) = -5.1, 90% CI 2-sided [-28.0 to 20.1]

16. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs), Serious Adverse Events (SAEs), Treatment Related AEs and SAEs
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included both SAEs and all non-SAEs. Treatment emergent AEs (TEAEs) were events that occurred between first dose of study drug and up to 4 weeks after last dose that were absent before treatment or that worsened relative to pretreatment state. A treatment-related AE was any untoward medical occurrence attributed to the study drug in a participant who received study drug. Relatedness to study drug was assessed by the investigator.
Time Frame: Day 1 of study drug dose to maximum of 4 weeks post last dose (maximum up to 16 weeks)
Population: Safety analysis set (SAS) included participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 37 | 37 | 37 | 36 | 37 | 49 | 36 | 36 | 38
Participants
  Treatment-emergent AEs | 17 | 16 | 14 | 17 | 14 | 20 | 13 | 18 | 12
  Treatment-emergent SAEs | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0
  Treatment-related AEs | 1 | 0 | 2 | 2 | 3 | 2 | 3 | 3 | 1
  Treatment-related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With TEAEs by Severity
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AE was assessed according to severity; mild (not causing any significant problem, dose adjustment not required), moderate (caused problem that does not interfere significantly with usual activities or the clinical status, dose adjustment needed due to adverse event) and severe (caused problem that interfered significantly with usual activities or the clinical status, study drug stopped due to adverse event).
Time Frame: Day 1 of study drug dose to maximum of 4 weeks post last dose (maximum up to 16 weeks)
Population: SAS included participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 37 | 37 | 37 | 36 | 37 | 49 | 36 | 36 | 38
Participants
  Mild | 12 | 9 | 11 | 11 | 7 | 8 | 7 | 11 | 6
  Moderate | 5 | 7 | 3 | 5 | 7 | 11 | 6 | 5 | 6
  Severe | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0

18. Secondary Outcome: Number of Participants Who Discontinued From Study Due to Adverse Events
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship.
Time Frame: Day 1 of study drug dose to maximum of 4 weeks post last dose (maximum up to 16 weeks)
Population: SAS included participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 37 | 37 | 37 | 36 | 37 | 49 | 36 | 36 | 38
Participants | 1 | 1 | 3 | 0 | 2 | 1 | 1 | 2 | 1

19. Secondary Outcome: Number of Participants With Laboratory Abnormalities Meeting Specified Criteria
Description: Bilirubin: greater than (>) 1.5* upper limit normal (ULN); aspartate aminotransferase, alanine aminotransferase: >2.5*ULN; creatinine, cystatin C: >1.3*ULN; creatine kinase: >2.0*ULN; glomerular filtration rate (GFR) CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration) Equat: less than (<) 60 milliliter (mL)/minute (min)/1.73 meter(m)^2, greater than or equal to (>=) 30% decrease from baseline; GFR: <60 mL/min/1.73m^2.
Time Frame: Day 1 of study drug dose to maximum of 4 weeks post last dose (maximum up to 16 weeks)
Population: SAS included participants who received at least 1 dose of investigational product. Here, 'overall number of participants analyzed' signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 37 | 36 | 36 | 36 | 37 | 49 | 35 | 36 | 38
Participants | 7 | 6 | 11 | 7 | 5 | 12 | 5 | 6 | 15

20. Secondary Outcome: Number of Participants With Categorical Summary of Post-Baseline Electrocardiogram (ECG) Data
Description: Following were ECG criteria used for categorical summary:1) PR interval: percentage change >=25/50%, QRS interval: value >140 msec, and QT interval corrected using the Fridericia's formula (QTcF): 450 msec < value less than equal to (<=) 480 and 30 < change <=60.
Time Frame: Post-baseline to Week 6, Post-baseline to Week 12
Population: SAS included participants who receive at least 1 dose of investigational product
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 37 | 37 | 37 | 36 | 37 | 49 | 36 | 36 | 38
Participants
  Post-baseline to Week 6: PR interval (>=25/50 percent) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Post-baseline to Week 6: QRS interval (>=140 msec) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Post-baseline to Week 6: QTcF interval (30< Change <=60) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Post-baseline to Week 12: PR interval (>=25/50 percent) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
  Post-baseline to Week 12: QRS interval (>=140 msec) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 0
  Post-baseline to Week 12: QTcF interval (450< Value <=480) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1
  Post-baseline to Week 12: QTcF interval (30 < Chg <= 60) | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1

21. Secondary Outcome: Number of Participants With Categorical Summary of Post-Baseline Vital Signs Data
Description: Following were the vital signs criteria: 1) Pulse rate: value <40 beats per min (bpm), value >120 bpm; 2) Sitting diastolic blood pressure (DBP): value <50 mmHg; change >=20 mmHg increase; change >=20 mmHg decrease; 3) Sitting systolic blood pressure (SBP): value <90 mmHg, change >=30 mmHg increase, change >=30 mmHg decrease; 4) Supine DBP: value <50 mmHg, change >=20 mmHg increase, change >=20 mmHg decrease; 5) Supine SBP: value <90 mmHg, change >=30 mmHg increase, change >=30 mmHg decrease.
Time Frame: Post-baseline to Week 12
Population: SAS included participants who receive at least 1 dose of investigational product. Here, 'overall number of participants analyzed' signifies number of participants evaluable for this outcome measure and 'number analyzed' signifies number of participants evaluable at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 35 | 34 | 33 | 33 | 34 | 47 | 32 | 36 | 34
Participants
  Pulse rate < 40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse rate >120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting DBP (<50 mmHg): number analyzed (Participants) | 3 | 11 | 5 | 5 | 6 | 5 | 8 | 6 | 5
  Sitting DBP (<50 mmHg) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting DBP (>=20 mmHg increase): number analyzed (Participants) | 3 | 11 | 5 | 5 | 6 | 5 | 8 | 6 | 5
  Sitting DBP (>=20 mmHg increase) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting DBP (>=20 mmHg decrease): number analyzed (Participants) | 3 | 11 | 5 | 5 | 6 | 5 | 8 | 6 | 5
  Sitting DBP (>=20 mmHg decrease) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting SBP (<90 mmHg): number analyzed (Participants) | 3 | 11 | 5 | 5 | 6 | 5 | 8 | 6 | 5
  Sitting SBP (<90 mmHg) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Sitting SBP (>= 30 mmHg increase): number analyzed (Participants) | 3 | 11 | 5 | 5 | 6 | 5 | 8 | 6 | 5
  Sitting SBP (>= 30 mmHg increase) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Sitting SBP (>=30 mmHg decrease): number analyzed (Participants) | 3 | 11 | 5 | 5 | 6 | 5 | 8 | 6 | 5
  Sitting SBP (>=30 mmHg decrease) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Supine DBP (<50 mmHg): number analyzed (Participants) | 32 | 25 | 29 | 29 | 28 | 42 | 25 | 31 | 31
  Supine DBP (<50 mmHg) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine DBP (>= 20mmHg increase): number analyzed (Participants) | 32 | 25 | 29 | 29 | 28 | 42 | 25 | 31 | 31
  Supine DBP (>= 20mmHg increase) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 2
  Supine DBP (>=20 mmHg decrease): number analyzed (Participants) | 32 | 25 | 29 | 29 | 28 | 42 | 25 | 31 | 31
  Supine DBP (>=20 mmHg decrease) | 0 | 2 | 0 | 0 | 1 | 4 | 0 | 0 | 0
  Supine SBP (<90 mmHg): number analyzed (Participants) | 32 | 25 | 29 | 29 | 28 | 42 | 25 | 31 | 31
  Supine SBP (<90 mmHg) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Supine SBP (>=30 mmHg increase): number analyzed (Participants) | 32 | 25 | 29 | 29 | 28 | 42 | 25 | 31 | 31
  Supine SBP (>=30 mmHg increase) | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 2 | 1
  Supine SBP (>= 30 mmHg decrease): number analyzed (Participants) | 32 | 25 | 29 | 29 | 28 | 42 | 25 | 31 | 31
  Supine SBP (>= 30 mmHg decrease) | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1

22. Secondary Outcome: Number of Participants Classified Per Skin Tolerability Assessment Severity Grades on Day 1, Week 1, 2, 4, 6, 8, 10, 12, 14, 16
Description: At the site of study drug application, skin tolerability was assessed for non-lesional skin surrounding the plaques on a scale from 0 to 4. Grade 0= none (no evidence of local intolerance), Grade 1= mild (minimal erythema and/or edema, slight glazed appearance), Grade 2= moderate (definite erythema and/or oedema with peeling and/or cracking but needs no adaptation of posology), Grade 3= severe, reported as AE (erythema, oedema glazing with fissures, few vesicles or papules: consider removing topical agent [if still in place]), Grade 4= very severe, reported as AE (strong reaction spreading beyond the treated area, bullous reaction, erosions: removal of topical agent [if still in place]).
Time Frame: Day 1, Week 1, 2, 4, 6, 8, 10, 12, 14, 16
Population: SAS included participants who receive at least 1 dose of investigational product. Here, "number analyzed" signifies the number of participants evaluable at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
Number analyzed (Participants) | 37 | 37 | 37 | 36 | 37 | 49 | 36 | 36 | 38
Participants
  Day1: None | 36 | 37 | 36 | 36 | 36 | 48 | 35 | 36 | 37
  Day1: Mild | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
  Day1: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Day1: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day1: Very severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day1: Missing | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Week 1: number analyzed (Participants) | 36 | 36 | 37 | 36 | 37 | 49 | 36 | 36 | 37
  Week 1: None | 32 | 35 | 32 | 34 | 35 | 44 | 32 | 32 | 35
  Week 1: Mild | 1 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 1
  Week 1: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 1: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 1: Very severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 1: Missing | 3 | 1 | 4 | 0 | 2 | 4 | 4 | 2 | 1
  Week 2: number analyzed (Participants) | 35 | 36 | 36 | 36 | 36 | 48 | 35 | 36 | 37
  Week 2: None | 33 | 35 | 30 | 34 | 35 | 45 | 34 | 35 | 33
  Week 2: Mild | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 2
  Week 2: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Week 2: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2: Very severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 2: Missing | 1 | 1 | 5 | 1 | 1 | 2 | 0 | 1 | 2
  Week 4: number analyzed (Participants) | 34 | 34 | 34 | 35 | 35 | 47 | 32 | 35 | 35
  Week 4: None | 34 | 32 | 29 | 32 | 34 | 44 | 30 | 32 | 30
  Week 4: Mild | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 3
  Week 4: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4: Very severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 4: Missing | 0 | 2 | 5 | 1 | 1 | 2 | 2 | 3 | 2
  Week 6: number analyzed (Participants) | 33 | 32 | 32 | 35 | 31 | 44 | 31 | 35 | 32
  Week 6: None | 32 | 31 | 26 | 30 | 27 | 37 | 28 | 31 | 30
  Week 6: Mild | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Week 6: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6: Very severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 6: Missing | 1 | 1 | 5 | 4 | 3 | 7 | 3 | 4 | 2
  Week 8: number analyzed (Participants) | 32 | 32 | 33 | 35 | 31 | 41 | 29 | 34 | 32
  Week 8: None | 29 | 30 | 27 | 30 | 26 | 34 | 26 | 30 | 28
  Week 8: Mild | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Week 8: Moderate | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Week 8: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8: Very severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 8: Missing | 2 | 2 | 6 | 4 | 4 | 6 | 3 | 4 | 4
  Week 10: number analyzed (Participants) | 32 | 31 | 32 | 33 | 31 | 40 | 28 | 34 | 30
  Week 10: None | 29 | 30 | 24 | 29 | 27 | 34 | 24 | 27 | 26
  Week 10: Mild | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Week 10: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10: Very severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 10: Missing | 3 | 1 | 7 | 3 | 3 | 6 | 4 | 7 | 4
  Week 12: number analyzed (Participants) | 36 | 36 | 36 | 35 | 35 | 46 | 34 | 36 | 35
  Week 12: None | 33 | 32 | 30 | 31 | 30 | 43 | 30 | 32 | 29
  Week 12: Mild | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Week 12: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
  Week 12: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12: Very severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 12: Missing | 3 | 4 | 6 | 3 | 4 | 3 | 3 | 3 | 5
  Week 14: number analyzed (Participants) | 36 | 34 | 34 | 34 | 34 | 45 | 34 | 35 | 33
  Week 14: None | 31 | 27 | 24 | 29 | 30 | 34 | 26 | 26 | 28
  Week 14: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 14: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 14: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 14: Very severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 14: Missing | 5 | 7 | 10 | 5 | 4 | 11 | 8 | 9 | 5
  Week 16: number analyzed (Participants) | 35 | 35 | 35 | 35 | 32 | 45 | 34 | 35 | 33
  Week 16: None | 31 | 28 | 26 | 28 | 28 | 35 | 26 | 28 | 26
  Week 16: Mild | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Week 16: Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 16: Severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 16: Very severe | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 16: Missing | 4 | 7 | 9 | 7 | 4 | 10 | 8 | 6 | 7

ADVERSE EVENTS:
Time Frame: Day 1 of study drug dose to maximum of 4 weeks post last dose (maximum up to 16 weeks)
Description: Same event may appear as both an AE and a serious AE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. SAS included participants who received at least 1 dose of investigational product.
Arm/Group | Vehicle Once Daily (QD) | PF-06700841 0.1% QD | PF-06700841 0.3% QD | PF-06700841 1.0% QD | PF-06700841 3.0% QD | Pooled Vehicle BID | PF-06700841 0.3% BID | PF-06700841 1.0% BID | PF-06700841 3.0% BID
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/37 | 0/37 | 0/36 | 0/37 | 1/49 | 0/36 | 0/36 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/37 | 0/37 | 0/37 | 1/36 | 0/37 | 1/49 | 1/36 | 2/36 | 0/38
Other Adverse Events (participants affected / at risk) | 7/37 | 7/37 | 7/37 | 9/36 | 8/37 | 10/49 | 4/36 | 10/36 | 2/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Once Daily (QD) (N=37) | PF-06700841 0.1% QD (N=37) | PF-06700841 0.3% QD (N=37) | PF-06700841 1.0% QD (N=36) | PF-06700841 3.0% QD (N=37) | Pooled Vehicle BID (N=49) | PF-06700841 0.3% BID (N=36) | PF-06700841 1.0% BID (N=36) | PF-06700841 3.0% BID (N=38)
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombophlebitis septic (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspiration bursa (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle Once Daily (QD) (N=37) | PF-06700841 0.1% QD (N=37) | PF-06700841 0.3% QD (N=37) | PF-06700841 1.0% QD (N=36) | PF-06700841 3.0% QD (N=37) | Pooled Vehicle BID (N=49) | PF-06700841 0.3% BID (N=36) | PF-06700841 1.0% BID (N=36) | PF-06700841 3.0% BID (N=38)
Nasopharyngitis (Infections and infestations) | 4 | 3 | 1 | 6 | 3 | 3 | 1 | 7 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 2 | 1 | 0 | 2 | 2 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 0 | 2 | 2 | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 0 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from the study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/83/NCT03850483/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/83/NCT03850483/SAP_001.pdf